## STATISTICAL ANALYSIS PLAN

**PROTOCOL NO: HLAB-003** 

## Human Laboratory Study of ASP8062 for Alcohol Use Disorder Protocol Version No.: 6.0 Version Date: 13Jun2022

## **Study Sponsor:**

National Institute on Alcohol Abuse and Alcoholism

#### **Plan Authors:**

Charles B. Scott, Ph.D. Director of Biostatistics

Janet H. Ransom, Ph.D.
President
Fast-Track Drugs & Biologics, LLC
20010 Fisher Avenue, Suite G
Poolesville, MD, 20837

Daniel E. Falk, Ph.D.
Health Science Administrator
Division of Medications Development
National Institute on Alcohol Abuse and Alcoholism
National Institutes of Health
6700B Rockledge Dr
Bethesda MD 20892-6902

**Version Number 2.0** 

**Date:** 13 June 2022

NCT05096117

# **Table of Contents**

| 1. | ABBREVIATIONS1 | 11 |
|---|---|---|
| 2. | INTRODUCTION1 | 13 |
| 3. | PROTOCOL SUMMARY 1 3.1. Study Objectives 1 3.1.1. Primary 1 3.1.2. Secondary 1 3.2. Study Design 1 3.3. Study Endpoints 2 3.3.1. Primary Efficacy Endpoint 2 3.3.2. Secondary Efficacy Endpoints 2 3.3.3. Safety Endpoints 2 | 14<br>14<br>14<br>20<br>20<br>20 |
| 4 | 3.3.4. Compliance | |
| <ol> <li>4.</li> <li>5.</li> </ol> | ASSSESSMENT AND JUSTIFICATION OF STUDY ENDPOINTS | 23<br>23<br>23<br>23<br>24<br>24<br>24<br>25<br>er<br>25<br>25<br>25<br>26<br>27 |
| 6. | HYPOTHESES TO BE TESTED | 29 |
| 7. | SAMPLE SIZE CONSIDERATIONS | 30 |
| 8. | DATA QUALITY ASSURANCE | 31 |
| 9. | STATISTICAL CONSIDERATIONS 9.1. General Considerations 9.2. Participant Accountability and Protocol Deviations 9.3. Demographics and Other Baseline Characteristics 9.4. Efficacy Analysis 9.4.1. Primary Analysis of the Primary Efficacy Endpoint 9.4.2. Confirmatory Secondary Endpoints 9.4.3. Analysis of the Secondary Endpoints 9.4.3. Analysis of the Secondary Endpoints | 32<br>32<br>33<br>33<br>33 |

| | 9.4.3.1. | Secondary Drinking Endpoints | 34 |
|---|---|---|---|
| | 9.4.3.2. | Alcohol Consequences and Craving Scales | |
| | 9.4.3.3. | Smoking and Any Nicotine Use | |
| | 9.4.3.4. | Sleep and Mood Scales | |
| | | e Adjustment for the Analysis of Secondary Efficacy Endpoi | |
| | | Sing Data | |
| | | Events | |
| | | Laboratory and Point of Care Tests | |
| | | ns, ECG, and Body Weight | |
| | | AR Scores | |
| | | '-R Scores | |
| | | nd Retention Analyses | |
| | | Ad Hoc Analyses | |
| | | tifeia Scale | |
| | 9.9.2 Supplem | ental Exploratory Analysis | 37 |
| 10. | VALIDATION OF PRO | GRAMMING CODE | 38 |
| 11. | | | |
| 12. | | FIGURE SHELLS | |
| | | Disposition, Participation, Compliance | |
| | | aphic and Baseline Characteristics | |
| | | Efficacy Endpoint | |
| | | atory Secondary Efficacy Endpoints | |
| | | ry Efficacy Endpoints | |
| | • | nalyses | |
| | 12.3. Figures | | 141 |
| | | List of Tables | |
| Table 1: | Subject Disposition - All | Randomized Subjects | 42 |
| Table 2: | Exposure to Investigation | nal Products Using AICure Data – mITT Subjects | 44 |
| Table 3: | Total Exposure to Investi | igational Products Using AICure Data – Evaluable Subjects. | 44 |
| Table 4: | Compliance to Investigat | ional Products Using AICure Data – mITT Subjects | 45 |
| Table 5: | Compliance to Investigat | ional Products Using AICure Data – Evaluable Subjects | 45 |
| Table 6: | AiCure Interventions mI | TT Subjects | 45 |
| Table 7: | AiCure Interventions – | Evaluable Subjects | 45 |
| Table 8: | • | nd Metabolite Plasma Levels – ASP8062 Arm Only (mITT | 46 |
| Table 9: | Summary of ASP8062 Pl | lasma Levels – ASP8062 Arm Only (Evaluable Subjects) | 47 |
| Table 10: | AiCure Report of ASP80 | 62 Versus ASP8062 Plasma Levels – mITT Subjects | 47 |

| Table 11: | AiCure Report of ASP8062 Versus ASP8062 Plasma Levels – Evaluable Subjects | 47 |
|---|---|---|
| Table 12: | Exit Interview – mITT Subjects | 47 |
| Table 13: | Exit Interview – Evaluable Subjects | 48 |
| Table 14: | Dropouts by Treatment Group and Week - mITT Subjects | 49 |
| Table 15: | Number and Percent of Subjects Using Brief Drinking Questions after Discontinuing TLFB – mITT Subjects | |
| Table 16: | Demographic Characteristics - mITT Subjects | 51 |
| Table 17: | Demographic Characteristics – Evaluable Subjects | 51 |
| Table 18: | Screening Cue Reactivity – mITT Subjects | 52 |
| Table 19: | Screening Cue Reactivity – Evaluable Subjects | 56 |
| Table 20: | Psychiatric Baseline Characteristics – mITT Subjects | 57 |
| Table 21: | Medical History – mITT Subjects | 57 |
| Table 22: | Baseline POMS – mITT Subjects. | 58 |
| Table 23: | Baseline POMS – Evaluable Subjects | 59 |
| Table 24: | Baseline PSQI – mITT Subjects | 59 |
| Table 25: | Baseline PSQI – Evaluable Subjects | 60 |
| Table 26: | Baseline Drinking-related Behavior and Characteristics – mITT Subjects | 61 |
| Table 27: | Baseline Drinking-related Behavior and Characteristics – Evaluable Subjects | 62 |
| Table 28: | Baseline Drinking by TLFB – mITT Subjects | 62 |
| Table 29: | Baseline Drinking by TLFB – Evaluable Subjects | 64 |
| Table 30: | Baseline Alcohol-Related Craving, Consequences, Withdrawal and Hyperkatifeia – m<br>Subjects | |
| Table 31: | Baseline Alcohol-Related Craving, Consequences, Withdrawal and Hyperkatifeia – Evaluable Subjects | 67 |
| Table 32: | Baseline Other Substance Use – mITT Subjects | 67 |
| Table 33: | Baseline Other Substance Use – Evaluable Subjects | 68 |
| Table 34: | Week 3 Strength of Craving Scores – mITT Subjects | 70 |
| Table 35: | Week 3 Strength of Craving Scores – Evaluable Subjects | 71 |
| Table 36: | ANCOVA Strength of Craving - mITT Subjects | 71 |
| Table 37: | ANCOVA Strength of Craving – Evaluable Subjects | 72 |
| Table 38: | ANCOVA Strength of Craving (Difference Alcohol-Water) – mITT Subjects | 74 |
| Table 39: | ANCOVA Strength of Craving (Difference Alcohol-Water) - Evaluable Subjects | 74 |
| Table 40: | Drinking Makes Things Perfect Scores - mITT Subjects | 75 |

| Table 41: | Drinking Makes Things Perfect Scores – Evaluable Subjects | 76 |
|---|---|---|
| Table 42: | ANCOVA Drinking Makes Things Perfect - mITT Subjects | 76 |
| Table 43: | ANCOVA Drinking Makes Things Perfect - Evaluable Subjects | 77 |
| Table 44: | ANCOVA Drinking Makes Things Perfect (Difference Alcohol-Water) - mITT Subje | cts77 |
| Table 45: | ANCOVA Drinking Makes Things Perfect (Difference Alcohol-Water) – Evaluable Subjects | 78 |
| Table 46: | Drink Now Scores- mITT Subjects | 78 |
| Table 47: | Drink Now Scores – Evaluable Subjects | 79 |
| Table 48: | ANCOVA Drink Now - mITT Subjects | 79 |
| Table 49: | ANCOVA Drink Now – Evaluable Subjects | 80 |
| Table 50: | ANCOVA Drink Now (Difference Alcohol-Water) - mITT Subjects | 80 |
| Table 51: | ANCOVA Drink Now (Difference Alcohol-Water) – Evaluable Subjects | 80 |
| Table 52: | Turn Down Drink Scores – mITT Subjects | 80 |
| Table 53: | Turn Down Drink Scores – Evaluable Subjects | 80 |
| Table 54: | ANCOVA Turn Down Drink – mITT Subjects | 80 |
| Table 55: | ANCOVA Turn Down Drink - Evaluable Subjects | 81 |
| Table 56: | ANCOVA Turn Down Drink (Difference Alcohol-Water) - mITT Subjects | 81 |
| Table 57: | ANCOVA Turn Down Drink (Difference Alcohol-Water) – Evaluable Subjects | 81 |
| Table 58: | Average of Cue Scores – mITT Subjects | 81 |
| Table 59: | Average of Cue Scores – Evaluable Subjects | 81 |
| Table 60: | ANCOVA Average of Cue Scores – mITT Subjects | 81 |
| Table 61: | ANCOVA Average of Cue Scores – Evaluable Subjects | 81 |
| Table 62: | ANCOVA Average of Cue Scores (Difference Alcohol-Water) – mITT Subjects | 81 |
| Table 63: | ANCOVA Average of Cue Scores (Difference Alcohol-Water) – Evaluable Subjects | 81 |
| Table 64: | Beverage Liking Scores – mITT Subjects | 81 |
| Table 65: | Beverage Liking Scores – Evaluable Subjects | 81 |
| Table 66: | Percentage of Subjects No Heavy Drinking Days Weeks 3-6 - mITT Subjects | 83 |
| Table 67: | Percentage of Subjects with No Heavy Drinking Days Weeks 3-6 – Full Model Logist Regression (mITT) | |
| Table 68: | Percentage of Subjects Abstinent from Alcohol Weeks 3-6 – mITT Subjects | 84 |
| Table 69: | Percentage of Subjects Abstinent from Alcohol Weeks 3-6 – Full Model Logistic Regression (mITT) | 84 |
| Table 70: | WHO 1-Level Decrease in Alcohol Consumption (mITT) – Weeks 3-6 | 85 |

| Table 71: | WHO 1-Level Decrease in Alcohol Consumption (mITT) – Full Model, Logistic Regression, Weeks 2-5 | . 85 |
|---|---|---|
| Table 72: | WHO 2-Level Decrease in Alcohol Consumption (mITT) – Weeks 3-6 | . 86 |
| Table 73: | WHO 2-Level Decrease in Alcohol Consumption (mITT) – Full Model, Logistic Regression, Weeks 3-6 | . 86 |
| Table 74: | Percentage of Days Abstinent per Week (mITT) – Weeks 3-6 | . 86 |
| Table 75: | Percentage of Days Abstinent per Week (mITT) Full Model, Mixed Effects, Weeks 3- | -687 |
| Table 76: | Percentage of Heavy Drinking Days per Week (mITT) – Weeks 3-6 | . 88 |
| Table 77: | Percentage of Heavy Drinking Days per Week (mITT) – Full Model, Mixed Effects, Weeks 3-6 | . 88 |
| Table 78: | Percentage of Very Heavy Drinking Days per Week (mITT) – Weeks 3-6 | . 88 |
| Table 79: | Percentage of Very Heavy Drinking Days per Week (mITT) – Full Model, Mixed Effect Weeks 3-6 | |
| Table 80: | Drinks per Week (mITT) – Weeks 3-6 | . 88 |
| Table 81: | Drinks per Week (mITT) – Full Model, Mixed Effects, Weeks 3-6 | . 88 |
| Table 82: | Drinks per Drinking Day (mITT) – Weeks 3-6 | . 88 |
| Table 83: | Drinks per Drinking Day (mITT) – Full Model, Mixed Effects, Weeks 3-6 | . 88 |
| Table 84: | Mean Cigarettes Smoked Among Smokers (mITT) – Weeks 3-6 | . 88 |
| Table 85: | Mean Cigarettes Smoked Among Smokers (mITT) – Full Model, Mixed Effects, Weeks 6 | |
| Table 86: | PACS (mITT) – Weeks 3-6 | . 88 |
| Table 87: | PACS (mITT) – Full Model, Mixed Effects, Weeks 3-6 | . 88 |
| Table 88: | Percentage of Subjects Abstinent from Nicotine Use <sup>1</sup> Weeks 3-6 – Among Subjects that Used Nicotine Products at Baseline | |
| Table 89: | Percentage of Subjects Abstinent from Nicotine Use <sup>1</sup> Weeks 3-6 – Full Model Logistic Regression (Among Nicotine Users at Baseline) | |
| Table 90: | Percentage of Subjects Abstinent from Smoking Weeks 3-6 – Among Baseline Smokers | 90 |
| Table 91: | Percentage of Subjects Abstinent from Smoking Weeks 3-6 – Full Model Logistic Regression (Among Baseline Smokers) | . 90 |
| Table 92: | PSQI Scores – mITT Subjects | . 91 |
| Table 93: | PSQI Scores (mITT) – Full Model, Mixed Effects, Weeks 5 & 7 | . 91 |
| Table 94: | POMS Total Mood Disturbance Score – mITT | . 92 |
| Table 95: | POMS Total Mood Disturbance Score (mITT) – Full Model, Mixed Effects, Weeks 5 & | 792 |
| Table 96: | POMS Tension-Anxiety Score – mITT Subjects | . 94 |
| Table 97: | POMS Tension-Anxiety Score (mITT) – Full Model, Mixed Effects, Weeks 5 & 7 | . 94 |

| Table 98: | POMS Anger-Hostility Score – mITT Subjects |
|---|---|
| Table 99: | POMS Anger-Hostility Score (mITT) – Full Model, Mixed Effects, Weeks 5 & 7 94 |
| Table 100: | POMS Vigor-Activity Score – mITT Subjects |
| Table 101: | POMS Vigor-Activity Score (mITT) – Full Model, Mixed Effects, Weeks 5 & 794 |
| Table 102: | POMS Fatigue-Inertia Score – mITT Subjects |
| Table 103: | POMS Fatigue-Inertia Score (mITT) – Full Model, Mixed Effects, Weeks 5 & 794 |
| Table 104 | POMS Confusion-Bewilderment Score – mITT Subjects |
| Table 105: | POMS Confusion-Bewilderment Score (mITT) – Full Model, Mixed Effects, Weeks 5 & 79 |
| Table 106: | POMS Depression-Dejection Score – mITT Subjects |
| Table 107: | POMS Depression-Dejection Score (mITT) – Full Model, Mixed Effects, Weeks 5 & 794 |
| Table 108: | PROMIS Negative Consequences of Alcohol Scores – mITT Subjects |
| Table 109: | ANCOVA PROMIS Negative Consequences of Alcohol – mITT Subjects |
| Table 110: | Overall Summary of Adverse Events – Safety Subjects |
| Table 111: | Number and Percentage of Subjects with Adverse Events - Safety Subjects |
| Table 112: | Summary of Subjects with Adverse Events by Severity and Relationship – ASP8062 100 |
| Table 113: | Summary of Subjects with Adverse Events by Severity and Relationship – Placebo 101 |
| Table 114: | Number and Percentage of Subjects with Adverse Events by Maximum Severity - Safety Subjects |
| Table 115: | Number and Percentage of Subjects Adverse Events by Relatedness - Safety Subjects 102 |
| Table 116: | Number and Percentage of Subjects with Treatment-Related Adverse Events by Maximum Severity- Safety Subjects |
| Table 117: | Number and Percentage of Subjects with Adverse Events Occurring in >= 5% of Subjects in Any One Group - Safety Subjects |
| Table 118: | Number and Percentage of Subjects with Adverse Events Leading to Discontinuation of Study - Safety Subjects |
| Table 119: | Number and Percentage of Subjects with Adverse Events Leading to Discontinuation of Study Drug – Safety Subjects |
| Table 120: | CIWA-AR Score > 10 at Least Once During Treatment - Safety Subjects |
| Table 121: | Summary of Vital Signs and Body Weights – Safety Subjects |
| Table 122: | Summary of ECG Results - Safety Subjects |
| Table 123: | Summary of Blood Chemistries and Hematology – Safety Subjects |
| Table 124: | Summary of Urinalysis Continuous Data – Safety Subjects |
| Table 125: | Summary of Urine Glucose and Nitrites – Safety Subjects 108 |

| Table 126: | Summary of Urine Protein, Ketones, Billirubin, Leukocyte Esterace, and Blood – S<br>Subjects | - |
|---|---|---|
| Table 127: | Summary of Positive Urine Drug Tests, Preganancy Test or BAC > 0.02 Any Time the Study– Safety Subjects | _ |
| Table 128: | Frequency of Subjects with Suicidal Ideation Any Time During the Study – Safety Subjects | 111 |
| Table 129: | Return to Baseline ACQ-SF-R Scores – Safety Subjects | 111 |
| | List of Listings | |
| Listing 1: Su | ubject Disposition - All Subjects | 114 |
| Listing 2. En | nrollment and Randomization – All Consented Subjects | 115 |
| Listing 3: R | eason not Eligible – Screen Failures | 115 |
| Listing 4: Pr | otocol Deviations – Safety Subjects | 115 |
| Listing 5: Su | ubjects Excluded from the Efficacy Analysis or Evaluable Set | 117 |
| Listing 6: D | emographics Data – Safety Subjects | 118 |
| Listing 7: Ba | aseline Drinking Characteristics – mITT Subjects | 118 |
| Listing 8: Ba | aseline Smoking Characteristics – mITT Subjects | 119 |
| Listing 9: M | INI DSM-5 Disorders – Safety Subjects | 119 |
| Listing 10: N | MINI DSM-5 AUD – Safety Subjects | 120 |
| Listing 11: N | Medical History – Safety Subjects | 120 |
| Listing 12: I | Orinking Goal – mITT Subjects | 121 |
| Listing 13: I | Physical Exam – Safety Subjects | 121 |
| Listing 14: I | Daily and Weekly Standard Drink Units (TLFB) During Treatment – mITT Subjects | 122 |
| Listing 15: I | Brief Drinking Questionnaire – mITT Subjects | 122 |
| Listing 16: 0 | Cue Reactivity – mITT Subjects | 122 |
| Listing 17: I | Orinking Consequences and Craving Scores – mITT Subjects | 123 |
| Listing 18: I | Pittsburg Sleep Quality Index Scores – mITT Subjects | 123 |
| Listing 19: S | Smoking and Other Nicotine Use Data- mITT Subjects | 124 |
| Listing 20: N | MINI AUD– Safety Subjects | 125 |
| Listing 21. I | Exit Interview – mITT Subjects | 126 |
| Listing 22: I | Orug Exposure from AiCure- mITT Subjects | 127 |

| Listing 23: 1 | Drug Accountability – Safety Subjects | 127 |
|---|---|---|
| Listing 24: | Take Control – mITT Subjects | 127 |
| Listing 25: | Adverse Events – Safety Subjects | 129 |
| Listing 26: S | Serious Adverse Events – Safety Subjects | 129 |
| Listing 27: 1 | POMS Scores – mITT Subjects | 131 |
| Listing 28. | Columbia-Suicide Severity Scale – Safety Subjects | 132 |
| Listing 29: 1 | Blood Chemistries – Safety Subjects | 133 |
| Listing 30: I | Hematology – Safety Subjects | 134 |
| Listing 31: U | Urinalysis – Safety Subjects | 135 |
| Listing 32: U | Urinalysis Microscopy <sup>1</sup> – Safety Subjects | 136 |
| Listing 33: 1 | Pregnancy Test/Birth Control Data – Safety Subjects | 137 |
| Listing 34: 1 | Blood Alcohol Concentration – Safety Subjects | 138 |
| Listing 35. U | Urine Drug Screen – Safety Subjects | 138 |
| Listing 36: | Vital Signs and Body Weights- Safety Subjects | 139 |
| Listing 37. I | ECG – Safety Subjects | 139 |
| Listing 38. I | Prior and Concomitant Medications – Safety Subjects | 139 |
| Listing 39: 1 | Blood for Drug Concentrations – Safety Subjects | 140 |
| Listing 40: 0 | Comments – Safety Subjects | 140 |
| | List of Figures | |
| Figure 1: | Percentage of Subjects No Heavy Drinking Days Weeks 3-6 | 142 |
| Figure 2: | Percentage of Subjects Abstinent Weeks 3-6 | 142 |
| Figure 3: | Weekly Percentage of Subjects No Heavy Drinking Days (mITT) | 142 |
| Figure 4: | Weekly Percentage of Subjects Abstinent (mITT) | 142 |
| Figure 5: | Weekly Percentage WHO 1-Level Decrease in Alcohol Consumption (mITT) | 142 |
| Figure 6: | Weekly Percentage WHO 2-Level Decrease in Alcohol Consumption No Imputation (mITT) | 142 |
| Figure 7: | Percentage Days Abstinent per Week Least Squares Means – (mITT) | 142 |
| Figure 8: | Percent Heavy Drinking Days per Week Lease Squares Means -(mITT) | 142 |
| Figure 9: | Mean Drinks per Week Lease Squares Means – (mITT) | 142 |
| Figure 10: | Mean Drinks per Drinking Day by Week Least Squares Means – (mITT) | 142 |

| Figure 11: | Weekly Number of Cigarettes Smoked in Smokers Over Entire Treatment Period – | Least |
|---|---|---|
| | Squares Means (mITT) | 142 |
| Figure 12: | Clinical Chemistry, Urinalysis, and Hematology Values Over Time | 142 |

# 1. ABBREVIATIONS

| - ADDREVITIONS | |
|---|---|
| Abbreviation | Definition |
| ACQ-SF-R | Alcohol Craving Scale – Short Form |
| AE | Adverse event |
| AICc | Akaike Information Criterion corrected for finite samples |
| ALT | Alanine aminotransferase |
| ANCOVA | Analysis of covariance |
| AST | Aspartate aminotransferase |
| AUD | Alcohol Use Disorder |
| BAC | Blood alcohol concentration |
| CI | Confidence interval |
| CIWA-AR | Clinical Institute Withdrawal Assessment for Alcohol-revised |
| CrCl | Creatinine clearance |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| CTCAE | Common terminology criteria for adverse events |
| dL | Deciliter |
| DSM-5 | Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| EDMS | Electronic Data Management System |
| EOS | End of study |
| F | Fahrenheit |
| FDA | Food and Drug Administration |
| g | Gram |
| GGT | Gamma-glutamyl transferase |
| hr | Hour |
| ICH | International Conference on Harmonization |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram |
| μg | Microgram |
| min | Minutes |
| MINI | MINI Neuropsychiatric Interview |
| mITT | Modified intention-to-treat |
| mL | Milliliter |
| mm | Millimeter |
| NHDD | No heavy drinking days |
| NIAAA | National Institutes on Alcohol Abuse and Alcoholism |
| OZ | Ounce |
| PACS | Penn Alcohol Craving Scale |
| POMS | Profile of Mood State |

| Abbreviation | Definition |
|--------------|----------------------------------------------------------|
| PROMIS | Patient Reported Outcomes Measurement Information System |
| PSNHDD | Percentage of subjects with no heavy drinking days |
| PSQI | Pittsburg Sleep Quality Index |
| PT | Preferred term |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SDU | Standard drinking unit |
| SOC | System Organ Class |
| THC | Tetrahydrocannabinol |
| TLFB | Timeline followback |
| TSH | Thyroid-stimulating hormone |
| ULN | Upper limit of normal |
| VAS | Visual analog scale |
| WHO | World Health Organization |

#### 2. INTRODUCTION

This statistical analysis plan (SAP) for Protocol No. HLAB-003, "Human Laboratory Study of ASP8062 for Alcohol Use Disorder" describes and expands upon the analytical plan presented in the protocol.

This document contains all planned analyses, reasons and justifications for these analyses for all study data. This plan also includes sample tables, figures, and listings that will be populated. The SAP will follow the International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines as indicated in Topic E3 (Structure and Content of Clinical Study Reports), Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials). The structure and content of the SAP provides sufficient detail to meet the requirements identified by the FDA and ICH.

The following sources were used in preparation of this SAP:

- Protocol # HLAB-003, Protocol Version No.: 6.0; Version Date: 13 Jun 2022
- ICH Guidance Topics E9, E3 and E8

#### 3. PROTOCOL SUMMARY

## 3.1. Study Objectives

## **3.1.1. Primary**

The primary objective of this study is to evaluate the effects of ASP8062, 25 mg once a day and matched placebo, on alcohol cue-elicited alcohol craving during a human laboratory paradigm after 2 weeks of daily dosing among subjects with moderate to severe alcohol use disorder (AUD) as confirmed by the Diagnostic and Statistical Manual of Mental Disorders – Fifth Edition (DSM-5<sup>TM</sup>).

## 3.1.2. Secondary

Secondary objectives include evaluation of ASP8062, 25 mg once a day, and matched placebo on reduction of alcohol consumption, alcohol craving, cigarette smoking (among smokers) and nicotine use (among nicotine users), mood, sleep, alcohol use negative consequences, study retention, and safety and tolerability throughout the last 4 weeks of the treatment phase of the study.

## 3.2. Study Design

This study is a 2-arm, double-blind, randomized, placebo-controlled, parallel group, 3-site study designed to assess the effects of ASP8062 as compared with placebo on responses to in vivo alcohol cue exposure in the human laboratory setting. After signing informed consent, subjects will be screened for eligibility and have other baseline assessments. Screening is permitted over a 14-day period and most baseline assessments will be performed on the day of randomization. Assessments include alcohol breathalyzer test (before signing consent), medical history, physical examination, weight, vital signs, electrocardiogram (ECG), drinking history by the timeline follow-back (TLFB) method, Clinical Institute Withdrawal Assessment for Alcohol-revised (CIWA-AR), prior medication use, MINI neuropsychiatric interview, urine drug test, smoking quantity frequency and nicotine use interview, clinical laboratory tests including chemistry, hematology, medical urinalysis, alcohol craving responses during a baseline cue reactivity session, Columbia Suicide Severity Rating Scale (C-SSRS), drinking goal, Penn Alcohol Craving Scale (PACS), Pittsburg Sleep Quality Index (PSQI), PROMIS Alcohol Negative Consequences short form, Profile of Moods State (POMS), Hyperkatifeia Scale and confirmation that subjects are treatment seeking and desire a reduction or cessation of drinking. Women of child-bearing potential will have a pregnancy test.

If eligible for the study, 60 subjects will be randomized using a stratified permuted block randomization procedure with "clinical site" as the stratification variable in an approximate 1:1 ratio (targeting 30 subjects per group) to receive either ASP8062 25 mg once daily or matched placebo for 6 weeks.

Subjects will be seen in the clinic at screening, at randomization and 5 other times during the study. A final follow-up telephone interview will occur ~2 weeks after the end of study in-clinic visit. Two cue reactivity sessions will be conducted. The first will be during screening (named pretreatment session) and the second will be after two weeks of investigational product

administration at Study Week 3. During these cue sessions, subjects will be presented with water, followed by alcohol and will be asked to respond to 4 individual visual analog scales (VAS) items assessing alcohol craving and 1 item assessing beverage liking. Other assessments during the treatment period include TLFB, clinical laboratory tests, blood for serum levels of study drug for determining study drug compliance, vital signs, ECG, concomitant medications, CIWA-AR, C-SSRS, pregnancy test, male and female birth control methods, adverse events (AEs), PACS, smoking quantity/frequency, PSQI, and POMS. The end of study visit will include the other assessments performed during the treatment phase and an Exit Interview, PROMIS questionnaire, and a treatment referral.

Study assessments and procedures will be performed at the visits and time points outlined in the Schedule of Assessments (**Table 1**).

**Table 1:** Schedule of Assessments

| Study Phase | Screening | Screening Treatment | | | | | | Follow-up<br>Call |
|---|---|---|---|---|---|---|---|---|
| Clinic Visit # | 1 | 2 | 3 | 4 | 5 | 6 | 7 | |
| Study Week (Days) <sup>b</sup> | -2 to -1<br>(-14 to -1) | 1<br>(1 to 7) | 2<br>(8 to 14) | 3<br>(15 to 21) | 4<br>(22 to 28) | 5<br>(29 to 35) | 7<br>(43 to 49) | 9<br>(57 to 63) |
| Informed Consent | X | | | | | | | |
| Alcohol Breathalyzer | X | X | X | X | X | X | X | |
| Urine Drug Test <sup>c</sup> | X | X | X | X | X | X | X | |
| Locator Form | X | Update | Update | Update | Update | Update | Update | |
| Demographics | X | | | | | | | |
| Medical History | X | Update | | | | | | |
| Physical Exam | X | Update | | | | | | |
| Body Weight | X | | | | X | | X | |
| MINI | X | | | | | | | |
| C-SSRS | | X | X | X | X | X | X | |
| Clinical Chemistry <sup>d</sup> | X | | | | X | | X | |
| Hematology <sup>e</sup> | X | | | | X | | X | |
| Medical Urinalysis <sup>f</sup> | X | | | | X | | X | |
| Pregnancy Test | X | X | | | | | X | |
| Birth control methods (all subjects) | X | Update | Update | Update | Update | Update | Update | |

| Study Phase | Screening | | End of<br>Study <sup>a</sup> | Follow-up<br>Call | | | | |
|---|---|---|---|---|---|---|---|---|
| Clinic Visit # | 1 | 2 | 3 | 4 | 5 | 6 | 7 | |
| Study Week (Days) <sup>b</sup> | -2 to -1<br>(-14 to -1) | 1<br>(1 to 7) | 2<br>(8 to 14) | 3<br>(15 to 21) | 4<br>(22 to 28) | 5<br>(29 to 35) | 7<br>(43 to 49) | 9<br>(57 to 63) |
| Vital Signs <sup>g</sup> | X | X | X | X | X | X | X | |
| Eligibility Checklist | X | X | | | | | | |
| Drinking Goal | X | | | | | | | |
| ECG | X | | | | X | | X | |
| Prior and Concomitant Meds | X | X | X | X | X | X | X | X |
| CIWA-AR | X | X | X | X | X | X | X | X |
| Screening Cue Reactivity Session:<br>VAS Scales | X | | | | | | | |
| Randomization | | X (Day 1) | | | | | | |
| Blood for Drug Concentration | | | | | X | | X | |
| Drug compliance/ accountability/<br>Review AiCure | | Dispense<br>Day 1 | X | X | X | X | X | |
| AEs (open ended question) | | X | X | X | X | X | X | X |
| Brief Telephone Interview <sup>h</sup> | | once during<br>the week | once during<br>the week | As needed if the subject misses a clinic visit | | | | |
| Take Control | | X | X | X | Xi | X | X | |
| Treatment Cue Reactivity Session:<br>VAS Scales | | | | X | | | | |

| Study Phase | Screening | Treatment | | | | End of<br>Study <sup>a</sup> | Follow-up<br>Call | |
|---|---|---|---|---|---|---|---|---|
| Clinic Visit # | 1 | 2 | 3 | 4 | 5 | 6 | 7 | |
| Study Week (Days) <sup>b</sup> | -2 to -1<br>(-14 to -1) | 1<br>(1 to 7) | 2<br>(8 to 14) | 3<br>(15 to 21) | 4<br>(22 to 28) | 5<br>(29 to 35) | 7<br>(43 to 49) | 9<br>(57 to 63) |
| TLFB | X | X | X | X | X | X | X | |
| Brief Drinking Questionnaire | as needed | | | | | | | |
| Exit Interview | | | | | | | X | |
| ACQ-SF-R | 2X pre/post<br>cue session | | | 2X pre/post<br>cue session | | | | |
| PACS | | X | X | X | X | X | X | |
| Cigarette smoking quantity/frequency and nicotine use | | X | | | | X | X | |
| PSQI | | X | | | | X | X | |
| POMS | | X | | | | X | X | |
| PROMIS Alcohol Negative<br>Consequences | | X | | | | | X | |
| Hyperkatifeia Scale | | X | | | | | | |
| Treatment Referral | | | | | | | X | |
| Follow-Up Telephone Interview | | | | | | | | X |
| Final Subject Disposition | | | | | | | | X |

<sup>&</sup>lt;sup>a</sup> EOS - end of study. These assessments are to be done at Week 7 or if the subject discontinues early and agrees to a final clinic visit.

<sup>&</sup>lt;sup>b</sup> Within each study week, there should be a least two days elapsed since the visit in the prior week.

- <sup>c</sup> Test for opiates (i.e., morphine test), cocaine, amphetamines, methamphetamine, THC, buprenorphine, methadone, benzodiazepines, oxycodone, barbiturates, 3,4-methylenedioxy-methamphetamine (MDMA also known as ecstasy), and EtG.
- d Creatinine, urea nitrogen, total bilirubin, ALT, AST, alkaline phosphatase, GGT, albumin, total cholesterol, triglycerides, sodium, potassium, and chloride
- <sup>e</sup> Complete blood cell count including RBC, WBC, hemoglobin, hematocrit, and platelets.
- A dipstick urinalysis will be performed that tests for specific gravity, ketones, pH, protein, blood, glucose, nitrites, bilirubin, and leukocyte esterase. If the dipstick is positive for blood, leukocyte esterase, or protein, then a microscopic analysis will be performed at the discretion of the investigator.
- g Sitting blood pressure and heart rate.
- <sup>h</sup> Telephone calls after the Week 1 and 2 in clinic visits will collect AEs, concomitant medications, CIWA-AR, and give a drug compliance reminder. The call during Week 2 should be several days before the cue session to remind the subject of the planned visit.
- <sup>i</sup> Two modules will be viewed this week.

## 3.3. Study Endpoints

## 3.3.1. Primary Efficacy Endpoint

The primary efficacy endpoint is the "strength" of alcohol craving VAS score (item 1 below) upon presentation of the first alcohol cue at Week 2 – after one week of investigational product treatment.

Confirmatory secondary endpoints include the VAS score for the other 3 VAS scales (items 2 through 4 below) for the first alcohol cue and the average score of the 4 VAS craving items; and the difference score (alcohol craving VAS scores minus the water craving VAS score). The verage liking VAS item is also a confirmatory secondary endpoint. The 4 VAS craving items in the order of presentation are:

- 1. How strong is your craving to drink alcohol? note this is the primary efficacy endpoint.
- 2. Having a drink would make things just perfect.
- 3. If I could drink alcohol now, I would drink it.
- 4. It would be hard to turn down a drink right now.

The beverage liking item is: How much did you like the beverage just given to you?

## 3.3.2. Secondary Efficacy Endpoints

Secondary efficacy endpoints will be analyzed over the last 4 weeks of the treatment period of treatment.

- 1. Percentage of subjects with no heavy drinking days. A "heavy drinking day" is 4 or more drinks per drinking day for women and 5 or more drinks per drinking day for men.
- 2. Percentage of subjects abstinent from alcohol
- 3. Percentage of subjects with at least a WHO 2-level decrease in alcohol consumption
- 4. Percentage of subjects with at least a WHO 1-level decrease in alcohol consumption
- 5. Percentage of days abstinent per week
- 6. Percentage of heavy drinking days per week
- 7. Percentage of very heavy drinking days per week. A "very heavy drinking day" is 8 or more drinks per drinking day for women and 10 or more drinks per drinking day for men.
- 8. Weekly mean number of drinks per week
- 9. Weekly mean drinks per drinking day
- 10. Cigarettes smoked per week among smokers
- 11. Percentage of subjects with no nicotine use among those reporting nicotine use at baseline
- 12. Alcohol craving score (PACS)
- 13. Sleep quality (PSQI) score

- 14. Profile of Mood States (POMS) score
- 15. PROMIS Alcohol Negative Consequences Score

## 3.3.3. Safety Endpoints

- 1. Vital signs
- 2. Body weight
- 3. Clinical laboratory parameters
- 4. BAC by breathalyzer
- 5. Urine drug tests
- 6. AEs
- 7. ECG results
- 8. CIWA-AR scores
- 9. Frequency of subjects with suicidal ideation at any time during the treatment period (C-SSRS)
- 10. Concomitant medication use
- 11. ACQ-SF-SR score (pre- and post-cue response sessions)

## 3.3.4. Compliance

Compliance will be assessed using the AiCure smart phone application and by tablet counts of returned blister packs at regular clinic visits. In addition, blood will be collected to determine plasma levels of ASP8062 and its metabolites. Compliance will be calculated as the percentage of investigational products taken as prescribed and by the total amount of study drug consumed. Participation in study visits will be evaluated as the percentage of subjects with complete drinking data. Compliance determined by ASP8062 plasma levels will be reported as number and percentage of subjects with a level above the limit of detection at each time point.

#### 4. **DEFINITION OF ANALYSIS SETS**

The study analysis populations will consist of the following:

Modified Intention-to-Treat (mITT) Analysis Set: The mITT set is defined as subjects randomized to participate in the study that took at least one dose of investigational product and had a non-missing VAS craving primary endpoint.

**Evaluable Analysis Set:** The evaluable analysis set for the secondary endpoints is defined as those subjects randomized to the study who took at least 1 tablet per day for at least 80% of days in Weeks 1-6.

**Safety Analysis Set:** The safety analysis set includes all subjects who took at least one dose of investigational product.

The analysis of the primary and confirmatory efficacy endpoints will be conducted on both the mITT and evaluable analysis sets. All secondary endpoint analyses will be performed on the mITT set. Weekly percentage heavy drinking days, mean number of drinks per week, and PACS scores will also be performed on the evaluable analysis set. Safety analyses will be conducted on the safety analysis set.

#### 5. ASSSESSMENT AND JUSTIFICATION OF STUDY ENDPOINTS

## **5.1.** Alcohol Craving Visual Analog Scales

Alcohol craving in response to a water and typical alcohol beverage cue is assessed using 4 individual VAS items adapted from the ACQ (Singleton-1994).

The VAS craving scale items include in the following order:

- 1. How strong is your craving to drink alcohol?
- 2. Having a drink would make things just perfect.
- 3. If I could drink alcohol now, I would drink it.
- 4. It would be hard to turn down a drink right now.

Anchors (scores) for items 1, 3, and 4 are: Strongly Disagree (0) to Strongly Agree (20).

Anchors (scores) for question 2 are: None (0) to Extremely Strong (20).

There will be no imputation for missing values.

## 5.2. Alcohol Consumption Endpoints

## 5.2.1. Daily Quantity of Alcohol Consumption

Drinking will be assessed using the TLFB methodology and Form 90 structured assessment pattern chart. The TLFB is a semi-structured interview that provides estimates of the daily quantity of alcohol consumption during specified time periods. It uses a calendar prompt and a number of other memory aids (e.g., holidays, payday, and other personally relevant dates) to facilitate accurate recall of drinking or other drug use during the target period. The procedure has been widely used in clinical and research contexts. It has demonstrated adequate levels of reliability and validity when administered as an in-person interview, over the telephone, and when administered via computer (Carey-1997, Sobell et al-1988, Sobell et al-1996).

If a subject is withdrawn from the study early and is no longer participating in clinic visits or providing TLFB drinking data but is willing to be contacted by phone at the week most proximal to dropout, then they will be asked about any drinking and heavy drinking during the time since last contact. Phone calls will continue until the end of the treatment period, as deemed acceptable by the patient. The two questions cover whether the subject had any heavy drinking days or drinking days during the period covered and will be used to capture drinking data in the absence of individual daily TLFB drinking data.

## 5.2.2. Drinking Days

A drinking day is one calendar day in which the subject reported any alcohol consumption (i.e., > 0 standard drinking units [SDUs]). A standard drink contains approximately 0.6 fluid ounces (oz) of pure alcohol. The data given by the subjects on amount and type of alcoholic beverage(s) consumed will be converted to SDUs. Standard drink unit definitions are provided in **Table 2**.

#### Table 2: Standard Drink Unit Definitions

For Beer (~ 5% alcohol), the approximate number of SDUs in:

- 12 oz = 1.0
- 16 oz = 1.3
- 24 oz = 2.0
- 40 oz = 3.3

For malt liquor ( $\sim 7\%$  alcohol), the approximate number of SDUs in:

- 12 oz = 1.4
- 16 oz = 1.9
- 22 oz = 2.6
- 40 oz = 4.7

For table wine (~ 12% alcohol), the approximate number of SDUs in:

- 750 mL bottle = 25 oz = 5.0
- 5 oz glass = 1.0
- 10 oz glass = 2.0

For 80 proof spirits (~ 40% alcohol), or hard liquor, the approximate number of SDUs in:

- 1.5 oz (mixed drink) = 1.0
- 16 oz (pint) = 8.5
- 25 oz (a fifth) = 17.0
- 1.75 L (59 oz) = 39.0

## **5.2.3.** Very Heavy and Heavy Drinking Day

A very heavy drinking day is defined as 8 or more drinks per day for a woman, and 10 or more for men. A heavy drinking day is defined as a day with 5 or more drinks (SDUs) for males and 4 or more drinks (SDUs) for females.

## 5.2.4. Days at Risk

If a subject is being treated at an inpatient facility, is incarcerated, or otherwise under confinement, the days spent in under these conditions is considered a reduction in the days at risk for drinking and is deducted from the denominator in calculations of rates of drinking days.

# 5.2.5. Percentage of Subjects with No Heavy Drinking Days and Percentage of Subjects Abstinent from Alcohol

The percentage of subjects with no heavy drinking days is the number of subjects that have no heavy drinking days during the period of interest divided by the number of subjects with at least one day of non-missing drinking data during the period of interest, multiplied by 100.

The percentage of subjects abstinent from alcohol is calculated similarly, except the numerator is the number of subjects that have no drinking days during the period of interest.

# 5.2.6. Weekly Percentage of Heavy Drinking Days and Weekly Percentage of Days Abstinent

Weekly percentage of heavy drinking days is the number of heavy drinking days in a 7-day period divided by 7 then multiplied by 100. The TLFB permits capturing data in a subsequent visit if a visit is missed; however, if fewer than 7 days are observed then the denominator is the number of days observed in the 7-day period. At least 3 days in a week must be observed; otherwise, the week is considered missing.

Weekly percentage of days abstinent is similarly calculated by using the number of days abstinent instead of the number of heavy drinking days.

# 5.2.7. Weekly Mean Number of Drinks and Weekly Mean Number of Drinks per Drinking Day

Weekly mean number of drinks is the sum of SDUs calculated to the tenths over 7 calendar days divided by the number of days with non-missing data. The quotient is multiplied by 7. At least 3 days in a week must be observed; otherwise, the week is considered missing.

Weekly mean number of drinks per drinking days utilizes the same numerator, and the denominator is the number of days with greater than 0 SDUs. Weeks where all days within the week are abstinent are assigned a value of 0 for weekly drinks per drinking day.

## 5.2.8. World Health Organization Drinking Risk Categorical Scale

The WHO has developed a drinking risk categorical scale that can be used in a responder analysis approach to assess clinically relevant decreases in alcohol consumption (<u>Aubin et al-2015</u>). Two dichotomous endpoints will be analyzed: WHO 1-level and WHO 2-level decrease in alcohol consumption. The WHO 1-level and 2-level decrease endpoints are the percentage of subjects experiencing at least a 1-level or 2-level decrease in WHO levels of alcohol consumption, respectively, from the level at baseline (the period including the 28 days before screening) to the level during the last 4 weeks of the maintenance phase (Study Weeks 2-5). The WHO levels of average alcohol consumption per day are as follows:

| | Males | Females |
|----------------|------------|-----------|
| Low Risk | 1 to 40g | 1 to 20g |
| Medium Risk | 41 to 60g | 21 to 40g |
| High Risk | 61 to 100g | 41 to 60g |
| Very High Risk | 101+g | 61+g |

where 14g = 1 SDU (WHO-2000). In computing the alcohol consumption level, average drinks per day will be used, computed as the sum of all drinking in the 28 day period divided by the number of days with non-missing drinking data in that period. Abstinent subjects will be included in a separate "Abstinent" category. A subject must have at least 1 week of data during the last 4 weeks of the maintenance phase to be considered non-missing.

## 5.3. Alcohol-Related Craving, Consequences, and Withdrawal

Alcohol-related craving is measured using the ACQ-SF-R scale and PACS; alcohol-related consequences are measured using the PROMIS Alcohol Negative Consequences scale; and alcohol-related withdrawal is measured using the CIWA-AR scale. The PACS and PROMIS

Alcohol Negative Consequences are used as efficacy endpoints, while the ACQ-SF-R and CIWA-AR scales are safety endpoints.

The ACQ-SF-R contains 12-items adapted from the 47-item ACQ-NOW developed by <u>Singleton et al (1994)</u> to assess craving for alcohol among alcohol users in the current context (right now). Items 3, 8, and 11 are reverse keyed. A general craving index is derived by summing all items and dividing by 12. If an item is missing, then the number of items is reduced by the number missing, and the sum is only the sum of the answered items. At least 10 items must be endorsed for the general craving index of ACQ-SF-R to be considered non-missing (i.e., scored).

The PACS is a five-item self-administered instrument for assessing craving (Flannery-1999). Frequency, intensity, and duration of thoughts about drinking are assessed along with ability to resist drinking. The final item asks the responder to provide an average rating of his/her craving over the course of the past week. The questions on the PACS use descriptors coupled with numerical ratings ranging from 0 to 6. The items are summed for a total score.

PROMIS Alcohol Negative Consequences scale is for negative consequences from alcohol use. The short form of the PROMIS Alcohol Negative Consequences questionnaire will be used to assess outcomes of alcohol use over the past 30 days (<u>Pilkonis-2013</u>).

#### The 7 PROMIS items include:

- Drinking created problems between me and others
- I disappointed others when I drank
- I was unreliable after I drank
- Others complained about my drinking
- I used poor judgment when I drank
- I said or did embarrassing things when I drank
- I had trouble getting things done after I drank

Each item is rated on a 5 point scale including: Never (1), Rarely (2), Sometimes (3), Often (4), and Almost Always (5) for the past 30 days. A subject's total score is converted to a T-score using scoring table provided by NIH PROMIS.

The CIWA-AR modified telephone version is an adaptation for telephone administration of the CIWA-AR a brief 10-item measure used to provide a quantitative index of the severity of the alcohol withdrawal syndrome (Sullivan et al-1989). The CIWA-AR has been used both in clinical and research applications and has demonstrated both reliability and validity (Sellers et al-1992, Stuppaeck et al-1994). The total score is the sum of the individual item scores. Since this is an interview scale, no missing items are anticipated. A score  $\geq$  10 is considered an indication that the subject is undergoing alcohol withdrawal.

#### **5.4. Mood**

Mood will be measured with the POMS, while negative emotional state will be measured using an exploratory measure of hyperkatifeia.

The POMS measures dimensions of affect or mood (McNair and Heuchert-2005). It consists of 65 adjectives to which the subject responds according to a 5-point scale ranging from "not at all (0)" to "extremely (5)." Six subscale scores will be computed for items grouped as follows: Tension-Anxiety, Depression-Dejection, Anger-Hostility, Vigor-Activity, Fatigue-Inertia, and Confusion-Bewilderment. A Total Mood Disturbance score will also be computed which consists of the sum of Tension-Anxiety, Depression-Dejection, Anger-Hostility, Fatigue-Inertia, and Confusion-Bewilderment scores then subtracting the Vigor-Activity subscale score. A missing value within a subscale will be replaced by the average score of the answered items within the subscale; if 2 or more items within a subscale are missing then the entire subscale is missing (Macefield et al-2010).

Hyperkatifeia is defined as a greater intensity of negative emotional/motivational signs and symptoms during withdrawal from drugs of abuse in the withdrawal/negative affect stage of the addiction cycle (Koob-2021). Hyperkatifeia or negative emotional state is considered to be one of stages of addiction in the context of drug withdrawal (Koob and LeMoal-1997, Koob-2019). NIAAA has developed a 24-item self-report Hyperkatifeia Scale to capture negative emotionality after stopping alcohol drinking that will be assessed for the first time in this study of heavy drinkers with a diagnosis of moderate to severe AUD. The items address four measures associated with negative emotional state including stress/anxiety, depression, stress, irritable and pain.

One difference between this scale and other negative emotional state scales is the pain questions. Pain may be particularly important in AUD as there is a positive association between pain severity and a higher risk for AUD (<u>Lawton and Simpson-2009</u>, <u>Edlund et al-2013</u>). Also, physical pain appears to be a significant predictor of alcohol use and heavy alcohol use and relapse to drinking after a period of abstinence (<u>Larson et al-2007</u>, <u>Caldeiro et al-2008</u>, <u>Witkiewitz et al-2015</u>).

## 5.5. Sleep Quality

Sleep quality will be measured using the PSQI. The PSQI is a 19-item questionnaire (<u>Buysse et al-1989</u>). The addition of all the scores permits an analysis of the subject's overall sleep experience in the past 30 days. The lower the overall score, the better the person sleeps. A score ≥ 5 is indictive of a sleep disturbance. If any of the items is missing, then the entire form is missing for that evaluation (PSQI website).

## 5.6. Cigarette Smoking Quantity-Frequency and Nicotine Use Questionnaire

A smoking quantity frequency and nicotine use interview will include 3 questions to assess nicotine use via cigarette smoking or via other products during the study: 1) Over the past week, on how many days did you smoke cigarettes?; 2) On the days you smoked during the past week, how many cigarettes did you smoke on average?; and 3) Over the past week, on how many days did you use other nicotine products (ex. chew, cigars, cigarellos, e-cigarettes, vape, gum, patch, etc...)? At baseline subjects that answer "0" to question #1 are considered non-smokers for the study. Cigarettes per week is the answer to question #1 multiplied by the answer to question #2. At baseline, subjects who report smoking (question #1) or the use of other nicotine product (question #3) will be considered nicotine users. The responses to questions #1 and #3 will be

| used to calculate the percentage of subjects abstinent from nicotine use among nicotine users. No imputation for missing values will be used. |
|---|

#### 6. HYPOTHESES TO BE TESTED

## 6.1. Primary Efficacy Endpoint

Subjects treated with ASP8062 will report significantly lower VAS alcohol craving ratings in response to the *in vivo* alcohol cue during the treatment human laboratory cue session than placebo-treated subjects.

The hypotheses for the confirmatory secondary endpoints for the cue reactivity sessions are the same as for the primary endpoint.

## 6.2. Secondary Efficacy Endpoints

It is hypothesized that, during the last 4 weeks of the treatment period, ASP8062 as compared to the placebo, will:

- 1. Increase the percentage of subjects with no heavy drinking days. A "heavy drinking day" is 4 or more drinks per drinking day for women and 5 or more drinks per drinking day for men.
- 2. Increase the percentage of subjects abstinent from alcohol
- 3. Increase the percentage of subjects with at least a WHO 2-level decrease in alcohol consumption
- 4. Increase the percentage of subjects with at least a WHO 1-level decrease in alcohol consumption
- 5. Increase the percentage of days abstinent per week
- 6. Decrease the percentage of heavy drinking days per week
- 7. Decrease the percentage of very heavy drinking days per week
- 8. Decrease the weekly mean number of drinks per week
- 9. Decrease the weekly mean drinks per drinking day
- 10. Decrease the weekly mean cigarettes smoked per week among smokers
- 11. Increase the percentage of subjects abstinent from nicotine use among subjects who used any nicotine products in the week before randomization
- 12. Decrease the mean alcohol craving score (PACS)
- 13. Decrease the mean PSQI score
- 14. Decrease total mood disturbance (POMS)
- 15. Decrease in alcohol negative consequences (PROMIS)

## 7. SAMPLE SIZE CONSIDERATIONS

Analysis of covariance with clinical site and baseline cue as the covariates will be used to model the primary outcome – the VAS craving score for the alcohol cue. Statistical power was estimated using [PASS 13] with the following parameters. The treatment effect parameter—a maximal 3-point study drug-placebo difference on the strength of VAS craving in response to the alcohol cue—was obtained from Roberts (2017), which used a similar cue reactivity paradigm. The mean values on this outcome at Week 3 are assumed to be 11 for ASP8062 and 14 for placebo and a standard deviation between subjects of 4. Clinical site and the baseline VAS craving for the alcohol cue were assumed to have correlations of 0.13 and 0.39, respectively, with the primary outcome. These correlations, coupled with assumed standard deviations for site and baseline VAS craving for the alcohol cue of 0.82 and 4, respectively, yield explained variation of 26%. These assumptions, with a sample size of 30 subjects per arm (60 total subjects), provides 87% statistical power with a 0.05 two-sided significance level.

#### 8. DATA QUALITY ASSURANCE

Data quality assurance will start with training of clinical investigative staff on data collection and assessment procedures including a Manual of Operations that describes what data to collect and procedures for completion of eCRFs. Completed eCRFs will be reviewed by Fast-Track Drugs and Biologics clinical monitors on a regular basis throughout the trial by comparison against the source documents.

Study data will come from the eCRFs, TLFB spreadsheets, coded AEs, coded medical history, AiCure Drug Compliance system outputs, and PK drug levels from the PK lab spreadsheets. eCRFs for this study were created using an electronic data management system (EDMS) based on IBM clinical development system. eCRFs were created using an established data dictionary for each variable including the field name, field type, field attributes, and coding for variables. Range checks, alpha-numeric requirements, and null/not null parameters were programmed as applicable. The back end database application is Oracle. Data entered into the EDMS system will be reviewed by Fast-Track clinical monitors and data managers. If incomplete or inaccurate data are found, the data will be queried in the system for site staff to address. The site will resolve data inconsistencies and errors using the EDMS with full audit trail of corrections being maintained within the system. Corrections and changes to the data will be reviewed by Fast-Track clinical monitors and data managers. TLFB spreadsheets have a double data entry check system and additionally, Fast-Track staff will verify the data entries with the drinking calandar to verify the correct percentages of alcohol by volume. QA review of laboratory data outputs is the responsibility of the individual testing laboratories; however, Fast-Track staff will verify that there is a result reported for each specimen that was recorded in the database as being collected. Coded AEs and medical history terms will be cross checked by a second trained MedDRA coder.

Additional edit checks will be written to detect anomalies in the database. These checks will address inconsistencies (within visits, across visits), invalid/unusual values, missing values, and protocol violations. Edit checking will be validated on test data or actual clinical trial data. In addition to programmed edit checks, quality control examination of data will also be performed on reviews of data listings.

#### 9. STATISTICAL CONSIDERATIONS

#### 9.1. General Considerations

For descriptive purposes, dichotomous and categorical variables will be presented as number of observations and percentages; continuous variables will be given as means, standard deviations (SD), median, miniumum (min) and maximum(max). Statistical tests will be two-tailed at a 0.05 Type I error rate. P-values for the primary and secondary endpoints of < 0.05 will be considered statistically significant. Endpoint data will also be screened for outliers and skewness. Appropriate non-parametric tests will be used to compare treatment groups on continuous baseline characteristics that are not normally distributed. Continuous endpoint data that are not normally distributed will be transformed using either a square root, logarithmic, or inverse transformation, the selection of which is determined by skewness and kurtosis statistics with values closest to zero. Cohen's d will be used to calculate the effect size for means and Cohen's h or odds ratios will be used to calculate the effect size for proportions. Descriptive statistics – mean, SD, median, min and max – of all endpoint data will be provided for each assement point or summarized at each week for drinking endpoints. All data will be presented in listings.

## 9.2. Participant Accountability and Protocol Deviations

A summary will be prepared to show dropouts/retention over time in each group, along with the reason for early discontinuation. The number of missing observations will be presented between groups. Protocol deviations will be presented as summaries by type of deviation.

## 9.3. Demographics and Other Baseline Characteristics

Summaries of the characteristics of the subjects in each of the study groups at baseline will be prepared for the mITT, and evaluable analysis sets. Demographic characteristics (e.g., age, gender, race, and ethnicity) and other baseline characteristics, coded medical history terms, screening cue session VAS scale scores and ACQ-SF-R pre and post session score, mood scales (e.g., POMS total and subscale scores), Hyperkatifeia Scale scores, PSQI, and drinking goal, MINI AUD scores and other DSM-5 diagnoses will be summarized by treatment group for the mITT and evaluable subjects. Chi-square tests or t-tests will be used on baseline characteristics to test the hypothesis of effective randomization. Imbalance in any of these factors is an indication of ineffective randomization which may bias the results observed on any of the endpoints.

Baseline drinking parameters in the 28-days prior to the start of screening, will be summarized by treatment group for the mITT subjects. t-tests will be used for baseline drinking parameters to test the hypothesis of effective randomization. The number and percentage of subjects with mild, moderate and severe symptoms of AUD and summary statistics for total number of symptoms will also be presented.

The quantity of cigarettes smoked per week in the week prior to randomization will be presented for those subjects who reported any smoking. The numbers and percentages of subjects who report other nicotine product use at baseline, any nicotine use, and who test positive for THC will also be presented. Because smoking, any nicotine use, and positive THC are subsets and are not

controlled by randomization, balance across treatment groups will be assessed using t-test and chi-square tests.

Baseline drinking-associated consequences (CIWA-AR and PROMIS Alcohol Negative Consequences scores) and drinking-associated-craving (PACS) total score and subscales will be summarized in the tables. t-test will be used to test for balance across the treatment groups and evaluate the hypothesis of ineffective randomization.

Continuous variables will be summarized using means, standard deviations, medians, minimum, and maximum values. Categorical variables will be summarized using counts and percentages.

## 9.4. Efficacy Analysis

## 9.4.1. Primary Analysis of the Primary Efficacy Endpoint

Each subject will have an initial alcohol cue for "strength" of craving score from the VAS that is the primary endpoint. Analysis of covariance (ANCOVA) with the "strength" of alcohol craving value as the dependent variable and the pretreatment "strength" of alcohol craving score from the alcohol cue as an independent fixed effect. Treatment and clinical site will also be included as independent factors.

No imputation for missing endpoint data will be performed.

## 9.4.2. Confirmatory Secondary Endpoints

There are 3 additional VAS craving questions and a beverage liking question asked during the human lab session. Each of these questions will be analyzed in the same manner as listed in Section 9.4.1. An overall mean of the 4 VAS craving items will also be analyzed similarly for just the alcohol beverage cue. The difference between the alcohol cue and water cue for each VAS item will be computed at both the pre and post treatment time points. The difference values for each VAS item and the average difference will be analyzed similarly to the primary endpoint.

## 9.4.3. Analysis of the Secondary Efficacy Endpoints

Secondary efficacy endpoints will also be analyzed based on data collected during the last 4 weeks of the maintenance period (Weeks 3 through 6), including TLFB and other questionnaire data assessed at Week 7 that reflect data collected during this period. Note that the data collected at Week 7 reflect drinking and other questionnaire items that occurred during Week 6.

In general, every continuous secondary efficacy endpoint is analyzed using a repeated measures mixed effects model where subjects are random effects; factors and covariates are fixed effects. The analyses will be performed using SAS PROC MIXED procedure. The information criterion is requested from every mixed effects model. Subjects are treated as a class variable and not continuous. The week (Weeks 3 through 6), treatment group, and clinical site are also treated as class variables.

The primary analysis model for all continuous endpoints is:

• Appropriately transformed endpoint = treatment + week + treatment\*week + clinical site + baseline equivalent of endpoint + other covariates (identified in Section 9.4.4)

This model will also be created for the untransformed endpoint. The solution statement from SAS PROC MIXED is requested to provide the solution for the fixed effects parameters. A

REPEATED statement specifies that values are repeated each week and subjects are nested within treatment group. The covariance structure is specified.

The selection of the covariance structure is performed using a simple repeated mixed effects model that includes treatment group as the only fixed effect and subject nested within treatment group as the only random effect. The covariance structure for each continuous secondary endpoint is selected from autoregressive, compound symmetry, Toeplitz, and unstructured. The Akaike Information Criterion (AICc) corrected for a finite sample is obtained from each of the four models for the four possible covariance structures to determine model fit. The smallest (minimum) AICc associated with one of the covariance structure is selected and the difference for each of the other three covariance structures are calculated. A graph is produced of the model fit statistics and relative difference for the four possible covariance structures. The graphs across the continuous endpoints are compared to determine which covariance structure will be selected for all continuous endpoints or if one or more models need different covariance structures.

Results based on the primary analysis model and the model of the untransformed endpoint will be presented in tabular form. The overall least squares means and least square means for each time point along with the 95% confidence intervals (CI) will be presented for the untransformed endpoint only, while two-tailed p-values and Cohen's d will be presented for both the untransformed and transformed data. Inference and Cohen's d will be based upon the results using appropriately transformed data. Graphs of all secondary endpoints will be produced.

## 9.4.3.1. Secondary Drinking Endpoints

Percentage of days abstinent per week, percentage of subjects abstinent, percentage of heavy drinking days per week, percentage of very heavy drinking days, weekly mean number of drinks per week, and weekly mean number of drinks per drinking day will be analyzed using the mixed effects model specified in Section 9.4.3. Covariates for these models will be identified as in Section 9.4.4.

Percentage of subjects with a WHO 1-level decrease, and WHO 2-level decrease in alcohol consumption risk category will be analyzed during the last 4 weeks of the maintenance period (Weeks 2 through 5) using a logistic regression model. Covariates for the logistic regression will be identified as in Section 9.4.4. 2x2 contingency tables will report the WHO 1-level decrease, and WHO 2-level decrease along with Cohen's h, odds ratios and 95% CIs. The Wald statistic will be used to test for treatment differences.

No adjustment for multiple comparisons and no imputation will be used for these endpoints.

## 9.4.3.2. Alcohol Consequences and Craving Scales

The PACS is assessed weekly and will be analyzed similarly to the drinking endpoint (Section 9.4.3.1). PROMIS alcohol negative consequences scale is assessed at baseline and Study Week 7 which will be used for the secondary endpoint. Analysis of covariance will be used to analyze the PROMIS scale similarly to the primary endpoint (Section 9.4.1).

No imputation or multiplicity adjustment will be used for this endpoint.

## 9.4.3.3. Smoking and Any Nicotine Use

The mean number of cigarettes smoked in the past week is measured weekly. The sample is the mITT subjects who smoked at baseline. The data will be analyzed as described in Section 9.4.3. Covariates for this endpoint will be identified in Section 9.4.4. Amount of other nicotine products is not captured, only number of days of use of other nicotine products. The analysis of days of use in subjects using other nicotine products at baseline will use the same method as cigarettes smoked. In addition, 2 tables will examine the number of subjects that are abstinent from cigarettes and any nicotine product use. There will be one logistic regression, if there are sufficient number of subjects abstaining from nicotine use, with abstaining as the dependent variable and covariates as described in Section 9.4.4. No imputation will be used for these endpoints.

## 9.4.3.4. Sleep and Mood Scales

The PSQI total score, POMS 6 subscales and total disturbance score are continuous variables. The data will be analyzed as described in Section 9.4.3. Covariates for these models will be identified as in Section 9.4.4.

No imputation or multiplicity adjustment will be used for these endpoints.

## 9.4.4. Covariate Adjustment for the Analysis of Secondary Efficacy Endpoints

Covariates for continuous secondary efficacy endpoints include the baseline equivalent of the endpoint, clinical site, treatment, time and the treatment by time interaction. Additional covariates for the secondary efficacy endpoints may include baseline characteristics with a theoretical and/or empirical basis for a relationship with a particular secondary endpoint. Such characteristics may include, but are not limited to, drinking goal (stop drinking versus reduce drinking but not stop), age, and baseline alcohol craving scale total score. Prior to the unblinding of the data, matrices of correlations between these baseline characteristics and each of the secondary efficacy endpoints, pooled across blinded treatment assignment, will be produced (using Pearson for continuous variables, Spearman for categorical outcomes). Selection of baseline variables to include as covariates in the models will be based on consideration of the following criteria: at least modest correlation with outcome (i.e.,  $r \ge 0.20$ ) and clinical expertise. Each endpoint may have a unique set of covariates. Care is taken to only select a limited number of covariates such that the models are not over fitted.

Covariates for the dichotomous secondary endpoints, percentage of subjects abstinent, WHO 1-level risk category decrease, and WHO 2-level risk category decrease in alcohol consumption, will use phi correlation with dichotomous variables, chi-square statistic for categorical variables, and biserial correlation. Fewer covariates for the logistic regression may be used depending upon the number of events. If the number of events permits the inclusion of a baseline drinking covariate, the percentage of days abstinent will be used as the covariate for the percent subjects abstinent endpoint and the percent heavy drinking days will be used as the covariate for the percent subjects with no heavy drinking days endpoint; however, no baseline drinking covariate will be employed for the endpoint, percent subjects with a WHO decrease in alcohol consumption, as this endpoint already adjusts for baseline drinking in its calculation.

## 9.5. Handling of Missing Data

The primary endpoint of craving cannot be imputed; likewise, for the other craving questions given during the human lab session. Secondary endpoints analyzed with mixed effects or logistic regression models are capable of handling missing data, so no imputation will be utilized. PROMIS scores are analyzed using ANCOVA which cannot handle missing data; therefore, only subjects with an assessment during the treatment period will be used and no imputation.

## 9.6. Safety Analysis

#### 9.6.1. Adverse Events

AEs will be coded using the most recent version of the Medical Dictionary for Regulatory Activities (MedDRA) and will be grouped by system, organ, and class (SOC) and preferred term (PT) designation. The severity, frequency, and relationship of AEs to investigational product will be presented by SOC and PT groupings. Listings of each individual AE including start date, stop date, severity, relationship, outcome, and duration will be provided. Each AE (based on PT) will be counted once only for a given study subject. If the same AE occurred on multiple occasions, the highest severity will be assumed. Thus, study subjects are not counted multiple times in a given numerator in the calculation of frequencies for a specific AE. C-SSRS reports of suicidality or suicidal ideation will be reported as AEs and analyzed as AEs if the investigator determines after an interview with the subject, that the responses are consistent with suicidal ideation or attempt.

## 9.6.2. Clinical Laboratory and Point of Care Tests

For clinical laboratory data, descriptive statistics will be generated for all tests performed at screening and at each clinic visit. If a laboratory analysis is repeated, the last measurement performed prior to the clinic visit will be used in the summary statistics for that clinic visit. If an unscheduled clinical laboratory visit occurs prior to a scheduled visit that is missed due to dropout, then the unscheduled visit will be used in the summary statistics for the missed scheduled clinical visit. If an unscheduled clinical laboratory visit occurs between two scheduled clinical visits, then the data from the unscheduled visit only be presented in the listings and not in summary statistics. In addition, at each post-randomization clinic visit descriptive statistics for change from baseline will be generated. Laboratory values will be plotted as mean  $\pm$  standard error over time. All laboratory measurements will be presented in the listings.

Number and percentage of positive urine drug tests and pregnancy tests for screening visits and all treatment and follow-up visits will be tabulated. Results of all urine drug tests and pregnancy tests will be presented in the listings. The percentage of subjects with a positive urine drug test at any time post start of treatment will also be presented by test type and treatment group.

## 9.6.3. Vital Signs, ECG, and Body Weight

Vital signs will be presented as summary statistics and change from baseline. The percentage of ECG results considered abnormal and clinically significant will be provided. Body weight will be presented as summary statistics and change from screening. Vital signs, ECG results, and weight measurements for all visits will be presented in the listings.
#### 9.6.4. CIWA-AR Scores

The number and percentage of subjects who reported CIWA-AR scores  $\geq 10$  at any time after the start of dosing will be presented.

## 9.6.5. ACQ-SF-R Scores

Summary statistics for ACQ-SF-R raw scores prior to after each cue session will be presented. The number and percentage of subjects with a higher ACQ-SF-R score post each cue session will be provided by treatment group.

## 9.7. Drug Exposure and Retention Analyses

Drug exposure will be presented for each treatment group as the mean number of tablets taken by week and overall through AiCure during the entire treatment phase. The analysis will include the total number of tablets taken and the percent compliance. AiCure data will also be used for the number subjects receiving reminder intervention (phone calls, texts, or in person visits). Compliance will also be evaluated by determining the proportion of subjects who were prescribed ASP8062, reported taking ASP8062 (by AiCure assessment), and had a plasma sample with detectable ASP8062. Compliance by ASP8062 plasma levels will be reported as number and percentage of subjects with a level above the limit of detection at each time point. Descriptive statistics of plasma levels of ASP8062 and metabolites will also be provided. Samples with levels below of limit of quantitation will not be included in the summary statistics and the N will reflect the number with a detectable level at each timepoint.

The participation rate is the percentage of subjects with complete drinking data. Dropouts by week with cumulative percentages will be provided by treatment arm.

### 9.8. Blood Alcohol Content

The number and percentage of subjects at any clinic visit that have a BAC > 0 will be tabulated. All BAC measurements will be presented in the listings.

#### 9.9. Exploratory and Ad Hoc Analyses

## 9.9.1. Hyperkatifeia Scale

There is interest in exploring the use of a new Hyperkatifeia Scale as a predictor of drug response and possibly as an outcome measure. *Ad hoc* analyses will be performed on this scale as a planned part of exploring the utility of this scale including subscales and individual items. *Ad hoc* analyses may include: 1) examining the association between cue outcomes and naturalistic outcomes; 2) conducting of moderator analyses; and 3) examining the treatment goal assessment and its relationship between outcomes. The data from this study could be used for combined analyses with results of other studies conducted in the future.

## 9.9.2 Supplemental Exploratory Analysis

The exploratory analysis are defined as: Explore moderators of the treatment effect on primary and secondary outcomes. The exploratory endpoint will not be analyzed at the same time as the primary and secondary endpoints.

#### 10. VALIDATION OF PROGRAMMING CODE

All SAS codes used to generate tables and listings will be validated and reviewed before being finalized. The validation process will be used to determine that the numbers are produced by a statistically valid method and that the execution of the computations is correct. Qualified personnel who have not previously been involved in the production of the original programming codes will perform the validation procedures. Methods of validation include independent programming and comparison to data listings. Tables will be reviewed for accuracy, consistency with this plan, consistency within tables, and consistency with corresponding output. Once validation is complete, a quality control reviewer will perform a final review of the documents for accuracy and consistency. Upon completion of validation and quality review procedures, all documentation will be collected and filed in the study documentation files at Fast-Track.

#### 11. REFERENCES

Aubin HJ, Reimer J, Nutt DJ, Bladstrom A, Torup L, Francois C, Chick J. Clinical relevance of as-needed treatment with nalmefene in alcohol dependent patients. Eur Addict Res. 2015;21:160–68.

Buysse, D. J., Reynolds, C. F., 3rd, Monk, T. H., et al. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989;28:193-213.

Caldeiro RM, Malte CA, Calsyn DA, Baer JS, Nichol P, Kivlahan DR, Saxon AJ. The association of persistent pain with out-patient addiction treatment outcomes and service utilization. Addiction. 2008;103:1996–2005.

Carey KB. Reliability and validity of the time-line follow-back interview among psychiatric outpatients: a preliminary report. Psych Addic Behav. 1997;11, 26-33.

Edlund MJ, Sullivan MD, Han X, Booth BM. Days with pain and substance use disorders: is there an association? Clin J Pain. 2013;29:689–695.

Flannery BA, Volpicelli JR, Pettinati HM. Psychometric properties of the Penn Alcohol Craving Scale. Alcohol Clin Exp Res 1999;23:1289-95.

Koob GF, Le Moal M. Drug abuse: hedonic homeostatic dysregulation. Science. 1997. 278:52–58.

Koob GF. Neurobiology of opioid addiction: opponent process, hyperkatifeia, and negative reinforcement. Biol Psychiatry. 2019;87:44–53.

Koob GF. Drug Addiction: Hyperkatifeia/Negative Reinforcement as a Framework for Medications Development. Pharmacol Rev. 2021;73:163-201.

Larson MJ, Paasche-Orlow M, Cheng DM, Lloyd-Travaglini C, Saitz R, Samet JH. Persistent pain is associated with substance use after detoxification: a prospective cohort analysis. Addiction. 2007;02:752–760.

Lawton J, Simpson J. Predictors of alcohol use among people experiencing chronic pain. Psychol Health Med. 2009:14:487–501.

Macefield RC, Metcalfe C, Lane JA, Donovan JL, Avery KNL, Blazeby JM, Down L, Neal DE, Hamdy FC, Vedhara K. Impact of prostate cance testing: evaluation of the emotional consequences of a negative biopsy result. Br J Cancer 2010;102:1335-1340.

Mason BJ, Light JM, Williams LD, Drobes DJ. Proof-of-concept human laboratory study for protracted abstinence in alcohol dependence: Effects of gabapentin. Addict Biol. 2009;14:73-83.

Mason BJ, Quello S, Goodell V, Shadan F. Gabapentin treatment for alcohol dependence. JAMA. 2014;174:70-77.

McNair DM, Heuchert JWP. Profile of Mood States (POMS) Multi-Health Systems, Tonawanda, NY. 2005.

Peduzzi P, Concato J, Kemper E, Holford TR, Feinstein AR. A simulation study of the number of events per variable in logistic regression analysis. 1996;49:1373-1379.

Pilkonis PA, Yu L, Colditz J, Dodds N, Johnston KL, Maihoefer C, Stover AM, Daley DC, McCarty D. Item banks for alcohol use from the Patient-Reported Outcomes Measurement Information System (PROMIS): use, consequences, and expectancies. Drug Alcohol Depend. 2013;130:167-77.

Roberts W, Harrison ELR, McKee S. Effects of varenicline on alcohol cue reactivity in heavy drinkers. Psychopharmacology (Berl). 2017;234:2737-2745.

Sellers EM, Sullivan JT, Somer G, Sykora K. Characterization of DSM-III-R criteria for uncomplicated alcohol withdrawal: proposal for a diagnostic inventory and revised withdrawal scale. In Naranjo, C. A. and Sellers, E. M. (Eds.) Novel pharmacological interventions for alcoholism. New York (pp. 369-71). 1992.

Singleton EG, Tiffany, ST, Henningfield JE. Development and validation of a new questionnaire to assess craving for alcohol. In: Harris LS (ed) *Problems of Drug Dependence, 1994; Proceedings of the 56<sup>th</sup> Annual Scientific Meeting, The College on Problems of Drug Dependence, Inc.* National Institute of Drug Abuse Research Monograph Series. Vol. 153. Rockville, MD 1995. p. 289.

Sobell LC, Sobell MB, Leo GI, Cancilla A. Reliability of a timeline method: assessing normal drinkers' reports of recent drinking and a comparative evaluation across several populations. Br J Addict. 1988;83:393-402.

Sobell LC, Brown J, Leo GI, Sobell MB. The reliability of the Alcohol Timeline Followback when administered by telephone and by computer. Drug Alcohol Depend 1996;42:49-54.

Stuppaeck CH, Barnas C, Falk M, Guenther V, Hummer M, Oberbauer H, Pycha R, Whitworth AB, Fleischhacker WW. Assessment of the alcohol withdrawal syndrome--validity and reliability of the translated and modified Clinical Institute Withdrawal Assessment for Alcohol scale (CIWA-A). Addiction. 1994;89:1287-92.

Sullivan JT, Sykora K, Schneiderman J, Naranjo CA, Sellers EM. Assessment of alcohol withdrawal: the revised clinical institute withdrawal assessment for alcohol scale (CIWA-AR). Br J Addict. 1989;84:1353-7.

Witkiewitz K, Maisto SA, Donovan DM. A comparison of methods for estimating change in drinking following alcohol treatment. Alcohol Clin Exp Res. 2010;34:2116–212.

World Health Organization (WHO): International Guide for Monitoring Alcohol Consumption and Related Harm. Geneva, WHO, 2000. Available at: http://whqlibdoc.who.int/hq/2000/who\_msd\_msb\_00.4.pdf.

- 12. TABLE, LISTING, AND FIGURE SHELLS
- **12.1.** Tables
- 12.1.1. Subject Disposition, Participation, Compliance

Table 1: Subject Disposition - All Randomized Subjects

| | ASP8062 | Placebo | Total | |
|---|---|---|---|---|
| | n (%) | n (%) | n (%) | p-value <sup>1</sup> |
| Number of Subjects Consented | | | XX | |
| Number of Subjects Screen Failed | | | XX | |
| Number of Subjects Randomized <sup>2</sup> | XX | XX | XX | 0.xxx |
| Number of Subjects Randomized not Receiving Study Drug | x (xx.x) | x (xx.x) | x (xx.x) | 0.xxx |
| Number of mITT Subjects | xx (xx.x) | xx (xx.x) | xxx (xx.x) | 0.xxx |
| Number of Completed <sup>3</sup> Subjects | xx (xx.x) | xx (xx.x) | xxx (xx.x) | 0.xxx |
| Number of Evaluable Subjects | xx (xx.x) | xx (xx.x) | xxx (xx.x) | 0.xxx |
| Number of Subject Completing Study & Drug | xx (xx.x) | xx (xx.x) | xx (xx.x) | 0.xxx |
| Number of Subjects Discontinuing Study Drug, Remaining in Study | xx (xx.x) | xx (xx.x) | xx (xx.x) | 0.xxx |
| Number of Subjects Withdrawn Early (did not provide any data at Week 7) | xx (xx.x) | xx (xx.x) | xx (xx.x) | 0.xxx |
| Reason for Early Withdrawal <sup>4</sup> | | | | |
| Subject withdrew consent | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Investigator withdrew subject | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Lost-to-followup | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Adverse Event | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Increased drinking | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Psychiatric crisis | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Died | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Absent from the protocol due to confinement in a controlled | xx(xx.x) | xx (xx.x) | xx (xx.x) | |
| environment | ( ) | | | |
| Determined after randomization to be ineligible | xx (xx.x) | xx (xx.x) | xx (xx.x) | |

Notes: <sup>1</sup> p-value from Fisher's exact test.

<sup>&</sup>lt;sup>2</sup>The following percentages are based upon number randomized

<sup>&</sup>lt;sup>3</sup>Completed is defined as attending all clinical visits through Week 7 making the subject available for all endpoint analyses

<sup>&</sup>lt;sup>4</sup>The following categories sum to the number of early withdrawals

Programmer Notes: The discontinuation reasons are as given on the CRF. Include only the reasons actually used for the subjects in the study. If a subject discontinued, but the specific reason is missing, include 'Missing' as a row in the table. Use the order of discontinuation reasons as presented on the CRF page.

**Table 2:** Exposure to Investigational Products Using AICure Data – mITT Subjects

| | Number of Tablets Taken | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | ASP8062<br>N=XX | | | | | Placebo<br>N=XX | | | |
| | N | Mean (SD <sup>3</sup> ) | Med | (Min-Max) | N | Mean (SD) | Med | (Min-Max) | p-value <sup>1</sup> |
| Week 1 | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | XX | xx.x (xx.x) | xx.x | (xx.x-xx.x) | 0.xxx |
| Week 2 | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | XX | xx.x (xx.x) | xx.x | (xx.x-xx.x) | 0.xxx |
| Week 3 | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | XX | xx.x (xx.x) | xx.x | (xx.x-xx.x) | 0.xxx |
| Week 4 | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | 0.xxx |
| Week 5 | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | 0.xxx |
| Week 6 | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | 0.xxx |
| Total Dose <sup>2</sup> | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | 0.xxx |

<sup>&</sup>lt;sup>1</sup> p-value from t-test

Table 3: Total Exposure to Investigational Products Using AICure Data – Evaluable Subjects

Same as Table 2 only using evaluable subjects

<sup>&</sup>lt;sup>2</sup> Dose is the total number of tablets taken, maximum prescribed is 42 tablets

<sup>&</sup>lt;sup>3</sup> SD is standard deviation

## Table 4: Compliance to Investigational Products Using AICure Data – mITT Subjects

Same analysis as Table 2 using compliance rather than dose. Compliance is the number of capsules taken/number of capsules prescribed.

## Table 5: Compliance to Investigational Products Using AICure Data – Evaluable Subjects

Same analysis as Table 4 using evaluable subjects

**Table 6:** AiCure Interventions mITT Subjects

| | | ASP8062 | Placebo | |
|----------------------------|----|-----------------|-------------------|----|
| | N | # Receiving ≥ 1 | N # Receiving ≥ 1 | |
| Interventions <sup>1</sup> | XX | XX | xx | XX |

<sup>&</sup>lt;sup>1</sup> Interventions includes texts, emails, and phone calls

## **Table 7:** AiCure Interventions – Evaluable Subjects

Same as Table 6 only using evaluable subjects

Table 8: Summary of ASP8062 and Metabolite Plasma Levels – ASP8062 Arm Only (mITT Subjects)

| | | ASP8062 | | |
|---|---|---|---|---|
| | N | % > LLD <sup>1</sup> | Mean (SD <sup>2</sup> ) | (Min-Max) |
| Week 4 | xx | xx.x | xx.x (xx.x) | (xx.x-xx.x) |
| Week 7 | xx | xx.x | xx.x (xx.x) | (xx.x-xx.x) |
| | | A | S3486189 | |
| | N | % > LLD <sup>1</sup> | Mean (SD <sup>2</sup> ) | (Min-Max) |
| Week 4 | xx | xx.x | xx.x (xx.x) | (xx.x-xx.x) |
| Week 7 | xx | xx.x | xx.x (xx.x) | (xx.x-xx.x) |
| | | A | S3486191 | |
| | N | % > LLD <sup>1</sup> | Mean (SD <sup>2</sup> ) | (Min-Max) |
| Week 4 | xx | xx.x | xx.x (xx.x) | (xx.x-xx.x) |
| Week 7 | xx | xx.x | xx.x (xx.x) | (xx.x-xx.x) |
| | | A | S3486192 | |
| | N | % > LLD¹ | Mean (SD <sup>2</sup> ) | (Min-Max) |
| Week 4 | xx | xx.x | xx.x (xx.x) | (xx.x-xx.x) |
| Week 7 | xx | xx.x | xx.x (xx.x) | (xx.x-xx.x) |

<sup>&</sup>lt;sup>1</sup> LLD is lowest level of detection<sup>2</sup> SD is standard deviation

Table 9: Summary of ASP8062 Plasma Levels – ASP8062 Arm Only (Evaluable Subjects)
Same as Table 8 only using evaluable subjects.

Table 10: AiCure Report of ASP8062 Versus ASP8062 Plasma Levels – mITT Subjects

| | | AiCure Report Indicates Drug Taken (pill count must = 1, on the day before the blood sample was drawn) | | | |
|---|---|---|---|---|---|
| Timing | Plasma level<br>Indicates Drug<br>Taken <sup>a</sup> | Yes, n (%) | No, n (%) | p-value <sup>b</sup> | kappa <sup>c</sup> |
| Week 4 | Yes | | | | |
| | No | | | | |
| Week 7 | Yes | | | | |
| | No | | | | |
| Overall | Yes | | | | |
| | No | | | | |

a Blood level of ≥xx ng/mL indicates drug taken

Table 11: AiCure Report of ASP8062 Versus ASP8062 Plasma Levels – Evaluable Subjects

Repeat of Table 10 using evaluable subjects

**Table 12:** Exit Interview – mITT Subjects

| ASP8062 | Placebo | Total |
|-----------|----------|-------|
| 1101 0002 | 1 Incebe | 1000 |

b Chi-square test for independence

c Kappa test for agreement

| Question | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
|---|---|---|---|---|
| D.1. 41.1 | | | | 0.xxx |
| Did you think you were receiving | | | | |
| the study drug or the placebo? | | | | |
| Placebo | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Study Drug | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Don't know; No idea | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| What is your desire to please | | | | 0.xxx |
| people? | | | | |
| More than average | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Average | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Less than average | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Take the study drug again, for | | | | 0.xxx |
| more than 6 weeks? | | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Did you ever miss a dose of | | | | |
| medication to avoid these effects? | | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Did you use any other services | | | | 0.xxx |
| during the study to help you | | | | |
| reduce drinking? | | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

<sup>&</sup>lt;sup>1</sup> p-value from chi-squared test (c) unless one of the cells expected is less than 5 then Fisher's exact test is used (f). Refuse to answer is not included in statistical test.

**Table 13:** Exit Interview – Evaluable Subjects

**Table 14:** Dropouts by Treatment Group and Week – mITT Subjects

| | | ASP8062<br>N=XX | | Placebo<br>N=XX | Total<br>N=XX | | |
|---|---|---|---|---|---|---|---|
| Study | | Cumulative | | Cumulative | | Cumulative | p-value <sup>1</sup> |
| Week <sup>2</sup> | n | n (%) | n | n (%) | n | n (%) | |
| Week 1 | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | 0.xxx |
| Week 2 | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | 0.xxx |
| Week 3 | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | 0.xxx |
| Week 4 | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | 0.xxx |
| Week 5 | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | 0.xxx |
| Week 6 | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | 0.xxx |
| Week 6 | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | 0.xxx |

<sup>&</sup>lt;sup>1</sup> Fisher's exact test

Table 15: Number and Percent of Subjects Using Brief Drinking Questions after Discontinuing TLFB – mITT Subjects

| | ASP8062 | Placebo | Total | |
|------------|-----------|---------|-------|----------------------|
| Study Week | n (%) | n (%) | n (%) | p-value <sup>1</sup> |
| Week 3 | xx (xx.x) | XX | XX.X | 0.xxx |
| Week 4 | XX | XX | XX.X | 0.xxx |
| Week 5 | XX | XX | XX.X | 0.xxx |
| Week 6 | XX | XX | XX.X | 0.xxx |
| Week 6 | XX | XX | XX.X | 0.xxx |
| Overall | XX | XX | XX.X | 0.xxx |

<sup>&</sup>lt;sup>1</sup>Fisher's exact test is used because frequencies are expected to be low

Note only rows with values above 0 will be presented

<sup>&</sup>lt;sup>2</sup>Subjects are considered dropouts when they stop providing TLFB and other data. Subjects that discontinue study drug but provide data are not considered dropouts.

**Demographic and Baseline Characteristics** 

12.1.2.

**Table 16: Demographic Characteristics - mITT Subjects** 

| Characteristic | ASP8062 | Placebo | Total | p-value <sup>1</sup> |
|---|---|---|---|---|
| Age (years) | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | xx.x | |
| $SD^2$ | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Gender | | | | 0.xxx |
| N | | | | |
| Male | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Female | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Race | | | | 0.xxx |
| N | XX | XX | XX | |
| White | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| African-American or Black | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Asian | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Native Hawaiian or Other Pacific Islander | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| American Indian or Alaskan Native | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Ethnicity | | | | 0.xxx |
| N | XX | XX | XX | _ |
| Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | _ |
| Not Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

¹c = chi-squared test, f=Fisher's exact test, w=Wilcoxon signed rank test

**Table 17:** Demographic Characteristics – Evaluable Subjects

<sup>&</sup>lt;sup>2</sup> SD is standard deviation

 Table 18:
 Screening Cue Reactivity – mITT Subjects

| | | | ASP8062 | Placebo | Total | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|
| | | | N=xx | N=xx | N=xx | |
| Cue | Question | Statistic | | | | |
| Water | Craving<br>Strength | | | | | 0.xxx |
| | | Mean (SD <sup>2</sup> ) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | xx | XX | XX | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| | Drinking makes things perfect | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | xx | xx | XX | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| | Drink now | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |

| | | | ASP8062<br>N=xx | Placebo<br>N=xx | Total<br>N=xx | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|
| | | Median | XX | XX | XX | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| | Turn down drink | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | XX | XX | XX | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| | Average | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | XX | XX | XX | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Alcohol | Craving<br>Strength | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | XX | XX | XX | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |

| | | ASP8062 | Placebo | Total | p-value <sup>1</sup> |
|---|---|---|---|---|---|
| | | N=xx | N=xx | N=xx | |
| Drinking makes things perfect | | | | | 0.xxx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | Median | XX | xx | XX | |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Drink now | | | | | 0.xxx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | Median | XX | xx | XX | |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Turn down drink | | | | | 0.xxx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | Median | XX | xx | XX | |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Average | | | | | 0.xxx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | Median | xx | XX | xx | |
| | | 1 | i e | 1 | |

| | | | ASP8062 | Placebo | Total | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|
| | | | N=xx | N=xx | N=xx | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Alcohol -<br>Water | Craving<br>Strength | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | XX | xx | XX | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| | Drinking makes<br>things perfect | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | XX | xx | XX | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| | Drink now | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | XX | xx | XX | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| | Turn down drink | | | | | 0.xxx |

| | | ASP8062<br>N=xx | Placebo<br>N=xx | Total<br>N=xx | p-value <sup>1</sup> |
|---|---|---|---|---|---|
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | Median | xx | XX | xx | |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Average | | | | | 0.xxx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | Median | xx | XX | xx | |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |

<sup>&</sup>lt;sup>1</sup> t-test is used to examine balance across treatment groups

 Table 19:
 Screening Cue Reactivity – Evaluable Subjects

<sup>&</sup>lt;sup>2</sup> SD is standard deviation

 Table 20:
 Psychiatric Baseline Characteristics – mITT Subjects

| | ASP8062 | Placebo | Total |
|------------------------|------------|------------|------------|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) |
| DSM-5 Disorders | | | |
| Depression | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Suicidality | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Manic | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Hypomanic | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Bipolar | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Panic | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Agoraphobia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Social Phobia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Obsessive Compulsive | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Posttraumatic Stress | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Substance Abuse | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Psychotic | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mood | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Anorexia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Bulemia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Binge-eating | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Generalized Anxiety | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Medical Organic | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Antisocial Personality | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

**Table 21:** Medical History – mITT Subjects

| | ASP8062 | Placebo | Total |
|---|---|---|---|
| Medical History SOC and Preferred Term | (N=xx) | (N=xx) | (N=xx) |
| SOC | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred term name | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

 Table 22:
 Baseline POMS – mITT Subjects

| | ASP8062 | Placebo | Total | p-value <sup>1</sup> |
|------------------------|---------|---------|---------|----------------------|
| Characteristic | (N=xx) | (N=xx) | (N=xx) | |
| Tension-Anxiety | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| $SD^2$ | xxx.xx | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Depression-Dejection | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | xxx.xx | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Anger-Hostility | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | xxx.xx | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Fatigue-Inertia | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | xxx.xx | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Confusion-Bewilderment | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | xx.x | XX.X | XX.X | |
| SD | xxx.xx | XXX.XX | XXX.XX | |

| | ASP8062 | Placebo | Total | p-value <sup>1</sup> |
|------------------------|---------|---------|---------|----------------------|
| Characteristic | (N=xx) | (N=xx) | (N=xx) | _ |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Vigor-Activity | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | xxx.xx | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Total Mood Disturbance | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | xxx.xx | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |

<sup>&</sup>lt;sup>1</sup> t-test

**Table 23:** Baseline POMS – Evaluable Subjects

**Table 24:** Baseline PSQI – mITT Subjects

| Characteristic | ASP8062 | Placebo | Total | p-value <sup>1</sup> |
|---|---|---|---|---|
| Overall Sleep Experience | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| $SD^2$ | xxx.xx | xxx.xx | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |

<sup>&</sup>lt;sup>2</sup>SD is standard deviation

| Characteristic | ASP8062 | Placebo | Total | p-value <sup>1</sup> |
|----------------|---------|---------|---------|----------------------|
| Scale Min-Max | | | (xx-xx) | |

#### **Table 25:** $Baseline\ PSQI-Evaluable\ Subjects$

<sup>&</sup>lt;sup>1</sup> t-test <sup>2</sup> SD is standard deviation

 Table 26:
 Baseline Drinking-related Behavior and Characteristics – mITT Subjects

| | ASP8062 | Placebo | Total | |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xx) | p-value <sup>1</sup> |
| Drinking Goal (n, %) | | | | |
| Stop Drinking | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Reduce but not stop | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Goal of no heavy drinking days (n, %) | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| # Drinks/Week Goal in Subjects that Want to | Reduce Drinking | | | |
| N | XX | XX | XX | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| $SD^2$ | XXX.XX | xxx.xx | xxx.xx | |
| Median | XX | XX | xx | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Motivation to achieve goal | | | | |
| N | XX | XX | XX | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | xxx.xx | xxx.xx | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Confidence in achieving goal | | | | |
| N | XX | xx | XX | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | xxx.xx | xxx.xx | |
| Median | XX | xx | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| AUD Symptom Severity (n, %) | | | | 0.xxx |
| Moderate (4 or 5 symptoms) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Severe (6 or more symptoms) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| AUD Number of Symptoms (n, %) | | | | |
| 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| 6 | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| 7 | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| 8 | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| 9 | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| 10 | xx (xx.x) | xx (xx.x) | xx (xx.x) | |

| | ASP8062 | Placebo | Total | |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xx) | p-value <sup>1</sup> |
| 11 | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| AUD Number of Symptoms (continuous) | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | xxx.xx | XXX.XX | |
| Median | XX | XX | XX | |

Note: Percentages are based on the number of non-missing values in each variable.

 Table 27:
 Baseline Drinking-related Behavior and Characteristics – Evaluable Subjects

**Table 28:** Baseline Drinking by TLFB – mITT Subjects

| | ASP8062 | Placebo | Total | |
|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Drinks/Week (Pre-screening Days -1 to -28) | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| $SD^2$ | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Drinks/Week (7 Days Prior to Randomization) | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |

<sup>1</sup> t-test

<sup>&</sup>lt;sup>2</sup>SD is standard deviation

| | ASP8062 | Placebo | Total | |
|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Drinks/Week (Percent Change Pre-screening Days | | | | 0.xxx |
| -1 to -28 to 7 Days Prior to Randomization) | | | | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Drinks/Drinking Day (Pre-screening Days -1 to - | | | | 0.xxx |
| 28) | | | | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Drinks/Drinking Day (7 Days Prior to | | | | 0.xxx |
| Randomization) | | | | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Drinks/Drinking Day (Percent Change Pre- | | | | 0.xxx |
| screening Days -1 to -28 to 7 Days Prior to | | | | |
| Randomization) | | | | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Percentage of Heavy Drinking Days | | | | 0.xxx |
| (Pre-screening Days -1 to -28) | | | | |
| Mean | xx.x% | xx.x% | xx.x% | |
| SD | xx.x% | xx.x% | xx.x% | |
| Median | xx.x% | xx.x% | xx.x% | |
| Min-Max | (xx%-xx%) | (xx%-xx%) | (xx%-xx%) | |
| Percentage of Very Heavy Drinking Days | | 1 | | 0.xxx |
| (Pre-screening Days -1 to -28) | | | | |
| Mean | xx.x% | xx.x% | xx.x% | |

| | ASP8062 | Placebo | Total | |
|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| SD | xx.x% | xx.x% | XX.X% | |
| Median | xx.x% | xx.x% | XX.X% | |
| Min-Max | (xx%-xx%) | (xx%-xx%) | (xx%-xx%) | |
| Percentage Days Abstinent | | | | 0.xxx |
| (Pre-screening Days -1 to -28) | | | | |
| Mean | xx.x% | xx.x% | XX.X% | |
| SD | xx.x% | xx.x% | XX.X% | |
| Median | xx.x% | xx.x% | XX.X% | |
| Min-Max | (xx%-xx%) | (xx%-xx%) | (xx%-xx%) | |
| WHO Risk Level | | | | 0.xxx |
| High Risk | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Very High Risk | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

Note: Percentages are based on the number of non-missing values in each variable.

**Table 29: Baseline Drinking by TLFB – Evaluable Subjects** 

<sup>&</sup>lt;sup>1</sup>Chi-square test for categorical variables and t-test for continuous variables <sup>2</sup> SD is standard deviation

Table 30: Baseline Alcohol-Related Craving, Consequences, Withdrawal and Hyperkatifeia – mITT Subjects

| | ASP8062 | Placebo | Total | |
|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Pre-cue ACQ-SF-R <sup>2</sup> | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| $SD^3$ | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx.x - xx.x) | |
| Post-cue ACQ-SF-R | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Pre-Post ACQ-SF-R | | | | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| PROMIS <sup>4</sup> Alcohol Negative | | | | 0.xxx |
| Consequences (T-scores) | | | | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| PACS <sup>5</sup> | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx.x - xx.x) | |
| CIWA-AR <sup>6</sup> | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx.x - xx.x) | |

| | ASP8062 | Placebo | Total | |
|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Withdrawal Symptoms (CIWA ≥ 10) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Hyperkatifeia | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | , , | , , , | (xx.x - xx.x) | |
| Stress Anxiety | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | , , | , , , | (xx.x - xx.x) | |
| Depression | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx.x - xx.x) | |
| Irritable | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx.x - xx.x) | |
| Pain | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx.x - xx.x) | |

<sup>&</sup>lt;sup>1</sup> t-test for continuous variables and chi-square test for categorical

<sup>&</sup>lt;sup>2</sup>ACQ-SF-R is Alcohol Craving Questionnaire – Short Form – Revised

<sup>&</sup>lt;sup>3</sup> SD is standard deviation

<sup>&</sup>lt;sup>4</sup> PROMIS is short form of Patient-reported Outcomes Information System

<sup>&</sup>lt;sup>5</sup> PACS is Penn Alcohol Craving Scale <sup>6</sup> CIWA-AR is Clinical Institute Withdrawal Assessment for Alcohol-revised

Table 31: Baseline Alcohol-Related Craving, Consequences, Withdrawal and Hyperkatifeia – Evaluable Subjects
Same as Table 30

**Table 32:** Baseline Other Substance Use – mITT Subjects

| | ASP8062 | Placebo | Total | |
|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Smoker (n, %) | xx (xx) | xx (xx) | xx (xx) | 0.xxx |
| Days Smoked in the Past Week | | | | |
| Mean | XX.X | XX.X | XX.X | |
| $SD^2$ | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| (Min-Max) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Average Cigarettes Smoked Per Week (among | | | | 0.xxx |
| Smokers) | | | | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Any Other Nicotine Product Use (doesn't include | xx (xx) | xx (xx) | xx (xx) | 0.xxx |
| cigarettes) (n, %) | | | | |
| Days Used Other Nicotine Products Per Week | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Any Nicotine Use (cigarettes + other) (n, %) | xx (xx) | xx (xx) | xx (xx) | 0.xxx |
| THC | | | | 0.xxx |
| Negative | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Positive | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

Note: Percentages are based on the number of non-missing values in each variable.

<sup>&</sup>lt;sup>1</sup>t-test for continuous variables and chi-square test for categorical

<sup>2</sup> SD is standard Deviation

**Table 33:** Baseline Other Substance Use – Evaluable Subjects

| 12.1.3. | Primary | <b>Efficacy</b> | <b>Endpoint</b> |
|---------|---------|-----------------|-----------------|

**Table 34:** Week 3 Strength of Craving Scores – mITT Subjects

| | | ASP8062 | Placebo | Total |
|---|---|---|---|---|
| | | N=xx | N=xx | N=xx |
| Cue | Statistic | | | |
| Water | | | | |
| | Mean (SD <sup>1</sup> ) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx | XX | XX |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) |
| Alcohol | | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx | XX | XX |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) |
| Alcohol - Water | | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx | XX | XX |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) |

<sup>&</sup>lt;sup>1</sup> SD is standard deviation

## **Table 35:** Week 3 Strength of Craving Scores – Evaluable Subjects

Same as Table 34

Table 36: ANCOVA Strength of Craving – mITT Subjects

## **Type III Wald Tests**

| Parameter | Num DF <sup>1</sup> | Den DF <sup>2</sup> | F Value | p-value |
|---|---|---|---|---|
| Arm | 1 | XX | xxx.xx | 0.xxx |
| Site | xx | xx | xxx.xx | 0.xxx |
| Baseline Cue <sup>3</sup> | 1 | XX | xxx.xx | 0.xxx |

<sup>&</sup>lt;sup>1</sup>Numerator degrees of freedom; <sup>2</sup> Demonimator degrees of freedom

# **Least Squares Means**

| | | | 95% CI | | | | | |
|---|---|---|---|---|---|---|---|---|
| Arm | Estimate | SE <sup>1</sup> | Lower CI | Upper CI | Difference | SE | p-value <sup>2</sup> | Cohen's d |
| ASP8062 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> Wald test;

<sup>&</sup>lt;sup>3</sup> Baseline Cue is the baseline equivalent of the outcome obtained after the presentation of the first alcohol cue at baseline

# Table 37: ANCOVA Strength of Craving – Evaluable Subjects

Follow the same analysis as Table 36
| 12.1.4. | Confirmatory Secondary Efficacy Endpoints |
|---------|-------------------------------------------|

Table 38: ANCOVA Strength of Craving (Difference Alcohol-Water) – mITT Subjects

Type III Wald Test

| Parameter | Num DF <sup>1</sup> | Den DF <sup>2</sup> | F Value | p-value |
|---|---|---|---|---|
| Arm | 1 | xx | xxx.xx | 0.xxx |
| Site | xx | xx | xxx.xx | 0.xxx |
| Baseline Cue <sup>3</sup> | 1 | xx | xxx.xx | 0.xxx |

<sup>&</sup>lt;sup>1</sup>Numerator degrees of freedom; <sup>2</sup> Demonimator degrees of freedom

#### **Least Squares Means**

| | | | 95% CI | | | | | |
|---|---|---|---|---|---|---|---|---|
| Arm | Estimate | SE <sup>1</sup> | Lower CI | Upper CI | Difference | SE | p-value <sup>2</sup> | Cohen's d |
| ASP8062 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> Wald test;

Table 39: ANCOVA Strength of Craving (Difference Alcohol-Water) – Evaluable Subjects

Same as Table 38

<sup>&</sup>lt;sup>3</sup> Baseline Cue is the baseline equivalent of the outcome obtained after the presentation of the first alcohol cue at baseline

 Table 40:
 Drinking Makes Things Perfect Scores – mITT Subjects

| | | ASP8062 | Placebo | Total |
|---|---|---|---|---|
| | | N=xx | N=xx | N=xx |
| Cue | Statistic | | | |
| Water | | | | |
| | Mean (SD <sup>1</sup> ) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx | XX | XX |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) |
| Alcohol | | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX | XX | XX |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) |
| Alcohol- Water | | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx | XX | xx |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) |

<sup>&</sup>lt;sup>1</sup> SD is standard deviation

**Table 41:** Drinking Makes Things Perfect Scores – Evaluable Subjects

Same as Table 40

Table 42: ANCOVA Drinking Makes Things Perfect – mITT Subjects

Type III Wald Test

| Parameter | Num DF <sup>1</sup> | Den DF <sup>2</sup> | F Value | p-value |
|---|---|---|---|---|
| Arm | 1 | xx | xxx.xx | 0.xxx |
| Site | 2 | xx | xxx.xx | 0.xxx |
| Baseline Cue <sup>3</sup> | 1 | xx | xxx.xx | 0.xxx |

<sup>&</sup>lt;sup>1</sup>Numerator degrees of freedom; <sup>2</sup> Demonimator degrees of freedom

## **Least Squares Means**

| | | | 95% CI | | | | | |
|---|---|---|---|---|---|---|---|---|
| Arm | Estimate | SE <sup>1</sup> | Lower CI | Upper CI | Difference | SE | p-value <sup>2</sup> | Cohen's d |
| ASP8062 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> Wald test;

<sup>&</sup>lt;sup>3</sup> Baseline Cue is the baseline equivalent of the outcome obtained after the presentation of the first alcohol cue at baseline

Table 43: ANCOVA Drinking Makes Things Perfect – Evaluable Subjects

Same analysis as Table 42

Table 44: ANCOVA Drinking Makes Things Perfect (Difference Alcohol-Water) – mITT Subjects

Type III Wald Test

| Parameter | Num DF <sup>1</sup> | Den DF <sup>2</sup> | F Value | p-value |
|---|---|---|---|---|
| Arm | 2 | xx | xxx.xx | 0.xxx |
| Site | 2 | xx | xxx.xx | 0.xxx |
| Baseline Cue <sup>3</sup> | 1 | xx | xxx.xx | 0.xxx |

<sup>&</sup>lt;sup>1</sup>Numerator degrees of freedom; <sup>2</sup> Demonimator degrees of freedom

#### **Least Squares Means**

| | | | 95% CI | | | | | |
|---|---|---|---|---|---|---|---|---|
| Arm | Estimate | SE <sup>1</sup> | Lower CI | Upper CI | Difference | SE | p-value <sup>2</sup> | Cohen's d |
| ASP8062 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> Wald test;

<sup>&</sup>lt;sup>3</sup> Baseline Cue is the baseline equivalent of the outcome obtained after the presentation of the first alcohol cue at baseline

Table 45: ANCOVA Drinking Makes Things Perfect (Difference Alcohol-Water) – Evaluable Subjects
Same analysis as Table 44

**Table 46:** Drink Now Scores-mITT Subjects

| | | ASP8062<br>N=xx | Placebo<br>N=xx | Total<br>N=xx |
|---|---|---|---|---|
| Cue | Statistic | | | |
| Water | | | | |
| | Mean (SD <sup>1</sup> ) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx | XX | xx |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) |
| Alcohol | | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx | XX | XX |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) |
| Alcohol - Water | | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |

| | ASP8062<br>N=xx | Placebo<br>N=xx | Total<br>N=xx |
|---------|-----------------|-----------------|---------------|
| Median | xx | xx | xx |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) |

<sup>&</sup>lt;sup>1</sup> SD is standard deviation

**Table 47: Drink Now Scores – Evaluable Subjects** 

Same as Table 46

**Table 48:** ANCOVA Drink Now – mITT Subjects

**Type III Wald Test** 

| Parameter | Num DF <sup>1</sup> | Den DF <sup>2</sup> | F Value | p-value |
|---|---|---|---|---|
| Arm | 1 | XX | xxx.xx | 0.xxx |
| Site | xx | xx | xxx.xx | 0.xxx |
| Baseline Cue <sup>3</sup> | 1 | xx | xxx.xx | 0.xxx |

<sup>&</sup>lt;sup>1</sup>Numerator degrees of freedom; <sup>2</sup> Demonimator degrees of freedom

<sup>&</sup>lt;sup>3</sup> Baseline Cue is the baseline equivalent of the outcome obtained after the presentation of the first alcohol cue at baseline

#### **Least Squares Means**

| | | | 95% CI | | | | | |
|---|---|---|---|---|---|---|---|---|
| Arm | Estimate | SE <sup>1</sup> | Lower CI | Upper CI | Difference | SE | p-value <sup>2</sup> | Cohen's d |
| ASP8062 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> Wald test;

**Table 49:** ANCOVA Drink Now – Evaluable Subjects

Same analysis as Table 48

Table 50: ANCOVA Drink Now (Difference Alcohol-Water) – mITT Subjects

Same analysis as Table 44 with difference as the dependent variable

**Table 51:** ANCOVA Drink Now (Difference Alcohol-Water) – Evaluable Subjects

Same analysis as Table 50

**Table 52:** Turn Down Drink Scores – mITT Subjects

Same analysis as Table 46

**Table 53:** Turn Down Drink Scores – Evaluable Subjects

Same analysis as Table 52

**Table 54:** ANCOVA Turn Down Drink – mITT Subjects

Same analysis as Table 48

**Table 55:** ANCOVA Turn Down Drink – Evaluable Subjects

Same analysis as Table 54

Table 56: ANCOVA Turn Down Drink (Difference Alcohol-Water) – mITT Subjects

Same analysis as Table 44

Table 57: ANCOVA Turn Down Drink (Difference Alcohol-Water) – Evaluable Subjects

Same analysis as Table 56

**Table 58:** Average of Cue Scores – mITT Subjects

Same analysis as Table 46

**Table 59:** Average of Cue Scores – Evaluable Subjects

Same as Table 58

**Table 60:** ANCOVA Average of Cue Scores – mITT Subjects

Same analysis as Table 48

**Table 61:** ANCOVA Average of Cue Scores – Evaluable Subjects

Same analysis as Table 60

Table 62: ANCOVA Average of Cue Scores (Difference Alcohol-Water) – mITT Subjects

Same analysis as Table 44

Table 63: ANCOVA Average of Cue Scores (Difference Alcohol-Water) – Evaluable Subjects

Same analysis as Table 62

**Table 64:** Beverage Liking Scores – mITT Subjects

Same analysis as Table 46

**Table 65:** Beverage Liking Scores – Evaluable Subjects

Same analysis as Table 64

| 12.1.5. | <b>Secondary</b> | <b>Efficacy</b> | <b>Endpoints</b> |
|---------|------------------|-----------------|------------------|
| | ~ ~ ~ ~ ~ ~ ~ , | | |

Table 66: Percentage of Subjects No Heavy Drinking Days Weeks 3-6 – mITT Subjects

| | ASP8062 | Placebo | Total |
|------------------------|------------|------------|------------|
| | (N=xx) | (N=xx) | (N=xxx) |
| No Heavy Drinking Days | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Table 67: Percentage of Subjects with No Heavy Drinking Days Weeks 3-6 – Full Model Logistic Regression (mITT)

| | | | | | | | | | 95% CI <sup>3</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF <sup>1</sup> | Estimate | Standard<br>Error | Wald<br>Chi-Square | Pr > Chi-<br>Square | Cohen's h | OR <sup>2</sup> | Upper | Lower |
| Intercept | | 1 | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | | | |
| Treatment | Overall | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | | | |
| Treatment <sup>4</sup> | ASP8062 | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | 0.xxx | xx.xxx | xx.xxx | xx.xxx |
| Site | Overall | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | | | |
| Site <sup>5</sup> | 1 | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | xx.xxx | xx.xxx | XX.XXX |
| Site | 2 | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | xx.xxx | xx.xxx | xx.xxx |

| | | | | | | | | 95% CI <sup>3</sup> | |
|---|---|---|---|---|---|---|---|---|---|
| Parameter | DF <sup>1</sup> | Estimate | Standard<br>Error | Wald<br>Chi-Square | Pr > Chi-<br>Square | Cohen's h | OR <sup>2</sup> | Upper | Lower |
| Cov | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | xx.xxx | XX.XXX | xx.xxx |

<sup>&</sup>lt;sup>1</sup> DF is degrees of freedom; <sup>2</sup> OR is odds ratio; <sup>3</sup> CI is confidence interval; <sup>4</sup> Comparison to placebo;

Programming note: COV is baseline equivalent of dependent variable and any other covariate(s) which have not been specified at the time of writing of SAP

#### Table 68: Percentage of Subjects Abstinent from Alcohol Weeks 3-6 – mITT Subjects

Presented in same manner as Table 66

# Table 69: Percentage of Subjects Abstinent from Alcohol Weeks 3-6 – Full Model Logistic Regression (mITT)

Prented in same manner as Table 67 programming note: baseline PDA is a covariate for PSA outcome

<sup>&</sup>lt;sup>5</sup> Site 3 is reference for the OR

Table 70: WHO 1-Level Decrease in Alcohol Consumption (mITT) – Weeks 3-6

| | ASP8062 | Placebo | Total |
|----------------------|------------|------------|------------|
| | (N=xx) | (N=xx) | (N=xxx) |
| WHO 1-Level Decrease | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Table 71: WHO 1-Level Decrease in Alcohol Consumption (mITT) – Full Model, Logistic Regression, Weeks 2-5

| | | | | | | | | | 95% CI <sup>3</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF <sup>1</sup> | Estimate | Standard<br>Error | Wald<br>Chi-Square | Pr > Chi-<br>Square | Cohen's h | OR <sup>2</sup> | Upper | Lower |
| Intercept | | 1 | xx.xxx | xx.xxx | XX.XXX | 0.xxx | | | | |
| Treatment | Overall | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | | | |
| Treatment <sup>4</sup> | ASP8062 | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | 0.xxx | xx.xxx | XX.XXX | XX.XXX |
| Site | Overall | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | | | |
| Site <sup>5</sup> | 1 | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Site | 2 | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | xx.xxx | XX.XXX | XX.XXX |
| Cov | | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | xx.xxx | xx.xxx | XX.XXX |

Programming note: COV is baseline equivalent of dependent variable and any other covariate(s) which have not been specified at the time of writing of SAP

Table 72: WHO 2-Level Decrease in Alcohol Consumption (mITT) – Weeks 3-6

Same as Table 70

Table 73: WHO 2-Level Decrease in Alcohol Consumption (mITT) – Full Model, Logistic Regression, Weeks 3-6

Same as Table 71

Table 74: Percentage of Days Abstinent per Week (mITT) – Weeks 3-6

| | | A | SP8062 | | | Placbo | | |
|---|---|---|---|---|---|---|---|---|
| Study<br>Week | N | Mean (SD <sup>1</sup> ) | Median | (Min-Max) | N | Mean (SD) | Median | (Min-Max) |
| 3 | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) |
| 4 | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) |
| 5 | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) |
| 6 | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) |
| Overall | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) |

<sup>&</sup>lt;sup>1</sup> SD is standard deviation

<sup>&</sup>lt;sup>1</sup> DF is degrees of freedom; <sup>2</sup> OR is odds ratio; <sup>3</sup> CI is confidence interval; <sup>4</sup> Comparison to placebo;

<sup>&</sup>lt;sup>5</sup> Site 3 is reference for the OR

Table 75: Percentage of Days Abstinent per Week (mITT) -- Full Model, Mixed Effects, Weeks 3-6

Type III Wald Tests

| Parameter | Num DF <sup>1</sup> | Den DF <sup>2</sup> | F Value | p-value |
|-----------|---------------------|---------------------|---------|---------|
| Arm | 1 | XXX | xxx.xx | 0.xxx |
| Week | 3 | XXX | xxx.xx | 0.xxx |
| Site | XX | XXX | xxx.xx | 0.xxx |
| Cov | X | XXX | xxx.xx | 0.xxx |
| Arm*Week | 5 | XXX | XXX.XX | 0.xxx |

<sup>&</sup>lt;sup>1</sup> Numerator degrees of freedom; <sup>2</sup> Denominator degrees of freedom

Programming note: Cov is the baseline equivalent of the dependent variable and any additional covariates included in the model.

#### **Least Squares Means**

| | | | | 95% | 6 CI <sup>2</sup> | | | Mo | odel |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE <sup>1</sup> | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d |
| ASP8062 | 3 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | 3 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| ASP8062 | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| ASP8062 | 5 | XX.XX | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | 5 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| ASP8062 | 6 | XX.XX | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | 6 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| ASP8062 | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |

Programming note: If a transformation of the dependent variable is used add 2 columns: p-value and Cohen's d for the transformed model.

Table 45 is the template for Tables 76, 78, 80, 82, 84, and 86. Table 75 is the template for Tables 77, 79, 81, 83, 85, and 87.

- Table 76: Percentage of Heavy Drinking Days per Week (mITT) Weeks 3-6
- Table 77: Percentage of Heavy Drinking Days per Week (mITT) Full Model, Mixed Effects, Weeks 3-6
- Table 78: Percentage of Very Heavy Drinking Days per Week (mITT) Weeks 3-6
- Table 79: Percentage of Very Heavy Drinking Days per Week (mITT) Full Model, Mixed Effects, Weeks 3-6
- Table 80: Drinks per Week (mITT) Weeks 3-6
- Table 81: Drinks per Week (mITT) Full Model, Mixed Effects, Weeks 3-6
- Table 82: Drinks per Drinking Day (mITT) Weeks 3-6
- Table 83: Drinks per Drinking Day (mITT) Full Model, Mixed Effects, Weeks 3-6
- Table 84: Mean Cigarettes Smoked Among Smokers (mITT) Weeks 3-6
- Table 85: Mean Cigarettes Smoked Among Smokers (mITT) Full Model, Mixed Effects, Weeks 3-6
- Table 86: PACS (mITT) Weeks 3-6
- Table 87: PACS (mITT) Full Model, Mixed Effects, Weeks 3-6

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> CI is confidence interval

Table 88: Percentage of Subjects Abstinent from Nicotine Use<sup>1</sup> Weeks 3-6 – Among Subjects that Used Nicotine Products at Baseline

| | ASP8062 | Placebo | Total |
|-----------------|------------|------------|------------|
| | (N=xx) | (N=xx) | (N=xxx) |
| No Nicotine Use | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

<sup>&</sup>lt;sup>1</sup> Nicotine use includes cigarettes or other nicotine products

Table 89: Percentage of Subjects Abstinent from Nicotine Use<sup>1</sup> Weeks 3-6 – Full Model Logistic Regression (Among Nicotine Users at Baseline)

| | | | | | | | | | 95% CI <sup>4</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF <sup>2</sup> | Estimate | Standard<br>Error | Wald<br>Chi-Square | Pr > Chi-<br>Square | Cohen's h | OR <sup>3</sup> | Upper CI | Lower CI |
| Intercept | | 1 | xx.xxx | xx.xxx | xx.xxx | 0.xxx | | | | |
| Treatment | Overall | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | | | |

| | | | | | | | | | 95% CI <sup>4</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF <sup>2</sup> | Estimate | Standard | Wald | Pr > Chi- | Cohen's h | OR <sup>3</sup> | Upper CI | Lower CI |
| | | | | Error | Chi-Square | Square | | | | |
| Treatment <sup>5</sup> | ASP8062 | X | xx.xxx | xx.xxx | xx.xxx | 0.xxx | 0.xxx | XX.XXX | xx.xxx | xx.xxx |
| Site | Overall | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | | | |
| Site <sup>6</sup> | 1 | X | xx.xxx | xx.xxx | xx.xxx | 0.xxx | | XX.XXX | xx.xxx | xx.xxx |
| Site | 2 | X | xx.xxx | xx.xxx | xx.xxx | 0.xxx | | XX.XXX | xx.xxx | xx.xxx |
| Cov | | X | xx.xxx | xx.xxx | xx.xxx | 0.xxx | | XX.XXX | xx.xxx | xx.xxx |

<sup>&</sup>lt;sup>1</sup> Nicotine use includes either cigarettes or other nicotine products; <sup>2</sup>DF is degrees of freedom; <sup>3</sup> OR is odds ratio; <sup>4</sup> CI is confidence interval; <sup>5</sup> Comparison to placebo for each active treatment; <sup>6</sup> Site 3 is reference for the OR

Programming note: COV is baseline equivalent of dependent variable and any other covariate(s) which have not been specified at the time of writing of SAP

Table 90: Percentage of Subjects Abstinent from Smoking Weeks 3-6 – Among Baseline Smokers

Same analysis as Table 88

Table 91: Percentage of Subjects Abstinent from Smoking Weeks 3-6 – Full Model Logistic Regression (Among Baseline Smokers)

Same analysis as Table 89

**Table 92:** PSQI Scores – mITT Subjects

| | | Λ. | SP8062 | | | | Placebo | |
|---|---|---|---|---|---|---|---|---|
| Study<br>Week | N | Mean (SD <sup>1</sup> ) | Median | (Min-Max) | N | Mean (SD) | Median | (Min-Max) |
| 1 | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) |
| 5 | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) |
| 7 | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) |

<sup>&</sup>lt;sup>1</sup> SD is standard deviation

Table 93: PSQI Scores (mITT) – Full Model, Mixed Effects, Weeks 5 & 7

Type III Wald Tests

| Parameter | Num DF <sup>1</sup> | Den DF <sup>2</sup> | F Value | p-value |
|---|---|---|---|---|
| Arm | 1 | XX | xxx.xx | 0.xxx |
| Site | xx | xx | xxx.xx | 0.xxx |
| Baseline PSQI | 1 | xx | xxx.xx | 0.xxx |

<sup>&</sup>lt;sup>1</sup> Numerator degrees of freedom; <sup>2</sup> Denominator degrees of freedom

# **Least Squares Means**

| | | | | 95% CI <sup>2</sup> | | | | Model | |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE <sup>1</sup> | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d |
| ASP8062 | 5 | XX.XX | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | 5 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| ASP8062 | 7 | XX.XX | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | 7 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> CI is confidence interval

Programming note: If a transformation of the dependent variable is used add 2 columns: p-value and Cohen's d for the transformed model.

**Table 94: POMS Total Mood Disturbance Score – mITT** 

| | | A | SP8062 | | Placebo | | | |
|---|---|---|---|---|---|---|---|---|
| Study<br>Week | N | Mean (SD <sup>1</sup> ) | Median | (Min-Max) | N | Mean (SD) | Median | (Min-Max) |
| 1 | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) |
| 5 | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) |
| 7 | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) |

<sup>&</sup>lt;sup>1</sup> SD is standard deviation

Table 95: POMS Total Mood Disturbance Score (mITT) – Full Model, Mixed Effects, Weeks 5 & 7

Type III Wald Tests

| Parameter | Num DF <sup>1</sup> | Den DF <sup>2</sup> | F Value | p-value |
|-----------|---------------------|---------------------|---------|---------|

| Parameter | Num DF <sup>1</sup> | Den DF <sup>2</sup> | F Value | p-value |
|-----------|---------------------|---------------------|---------|---------|
| Arm | 1 | xxx | xxx.xx | 0.xxx |
| Week | 1 | xxx | xxx.xx | 0.xxx |
| Site | 2 | xxx | xxx.xx | 0.xxx |
| Cov | X | xxx | xxx.xx | 0.xxx |
| Arm*Week | X | xxx | xxx.xx | 0.xxx |

<sup>&</sup>lt;sup>1</sup> Numerator degrees of freedom; <sup>2</sup> Denominator degrees of freedom

Programming note: Cov is the baseline equivalent of the dependent variable and any additional covariates included in the model.

## **Least Squares Means**

| | | | | 95% CI <sup>2</sup> | | | | Model | |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE <sup>1</sup> | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d |
| ASP8062 | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | 4 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| ASP8062 | 6 | XX.XX | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | 6 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| ASP8062 | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> CI is confidence interval

 $Programming\ note: If\ a\ transformation\ of\ the\ dependent\ variable\ is\ used\ add\ 2\ columns:\ p-value\ and\ Cohen's\ d\ for\ the\ transformed\ model.$ 

Table 94 is the template for Tables 96, 98, 100, 102, 104, and 106. Table 95 is the template for Tables 97, 99, 101, 103, 105, and 107

**Table 96: POMS Tension-Anxiety Score – mITT Subjects** 

Table 97: POMS Tension-Anxiety Score (mITT) – Full Model, Mixed Effects, Weeks 5 & 7

**Table 98: POMS Anger-Hostility Score – mITT Subjects** 

Table 99: POMS Anger-Hostility Score (mITT) – Full Model, Mixed Effects, Weeks 5 & 7

**Table 100:** POMS Vigor-Activity Score – mITT Subjects

Table 101: POMS Vigor-Activity Score (mITT) – Full Model, Mixed Effects, Weeks 5 & 7

**Table 102:** POMS Fatigue-Inertia Score – mITT Subjects

Table 103: POMS Fatigue-Inertia Score (mITT) – Full Model, Mixed Effects, Weeks 5 & 7

**Table 104 POMS Confusion-Bewilderment Score – mITT Subjects** 

Table 105: POMS Confusion-Bewilderment Score (mITT) – Full Model, Mixed Effects, Weeks 5 & 7

**Table 106:** POMS Depression-Dejection Score – mITT Subjects

Table 107: POMS Depression-Dejection Score (mITT) – Full Model, Mixed Effects, Weeks 5 & 7

**Table 108:** PROMIS Negative Consequences of Alcohol Scores – mITT Subjects

| | Placebo | | | | | | ANS-6637<br>200mg | |
|---|---|---|---|---|---|---|---|---|
| Study<br>Week | N | Mean (SD <sup>1</sup> ) | Median | (Min-Max) | N | Mean (SD) | Median | (Min-Max) |

| 1 | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) |
|---|----|----------|-----|---------|----|----------|-----|---------|
| 7 | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) |

<sup>&</sup>lt;sup>1</sup> SD is standard deviation

**Table 109:** ANCOVA PROMIS Negative Consequences of Alcohol – mITT Subjects

**Type III Wald Test** 

| Type III walu lest | | | | |
|---|---|---|---|---|
| Parameter | Num DF <sup>1</sup> | Den DF <sup>2</sup> | F Value | p-value |
| Arm | 1 | xx | xxx.xx | 0.xxx |
| Site | 2 | xx | xxx.xx | 0.xxx |
| <b>Baseline PROMIS</b> | 1 | xx | xxx.xx | 0.xxx |

<sup>&</sup>lt;sup>1</sup> Numerator degrees of freedom; <sup>2</sup> Demonimator degrees of freedom

## **Least Squares Means**

| | | | | 95% CI <sup>2</sup> | | | | Model | |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE <sup>1</sup> | Lower<br>CI | Upper CI | Difference | SE | p-value | Cohen's d |

| | | | | 95% CI <sup>2</sup> | | 95% CI <sup>2</sup> | | | Model |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE <sup>1</sup> | Lower<br>CI | Upper CI | Difference | SE | p-value | Cohen's d |
| ASP8062 | 7 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | 7 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> CI is confidence interval

Programming note: If a transformation of the dependent variable is used add 2 columns: p-value and Cohen's d for the transformed model.

# 12.1.6. Safety Analyses

**Table 110:** Overall Summary of Adverse Events – Safety Subjects

| | ASP8062 | Placebo | Total | |
|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Number of AEs | XX | XX | XX | |
| Number of SAEs | XX | XX | XX | |
| Number (%) of subjects with at least one AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Number (%) of subjects with at least one SAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Number (%) of subjects with at least one AE related <sup>2</sup> to study product | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Number of AEs by severity | | | | |
| Mild | XX | XX | XX | |
| Moderate | XX | XX | XX | |
| Severe | XX | XX | XX | |
| Life-threatening | XX | XX | XX | |
| Number of AEs by relationship to study product | | | | |
| At least possibly related | XX | XX | XX | |
| Unrelated | XX | XX | XX | |
| Number of AEs by SAE status | | | | |
| No | XX | XX | XX | |
| Yes | XX | XX | XX | |

<sup>&</sup>lt;sup>1</sup>p-value from chi-square test <sup>2</sup> Related is possible, probable, or definite

Table 111: Number and Percentage of Subjects with Adverse Events - Safety Subjects

| MedDRA System Organ Class/ | ASP8062 | Placebo |
|----------------------------|------------|------------|
| Preferred Term | (N=xx) | (N=xx) |
| - Any Adverse Events - | xx (xx.x%) | xx (xx.x%) |
| SOC | | |
| - Overall - | xx (xx.x%) | xx (xx.x%) |
| Preferred term 1 | xx (xx.x%) | xx (xx.x%) |
| Preferred term 2 | xx (xx.x%) | xx (xx.x%) |

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term.

Programmer's Notes: Order System Organ Class alphabetically and preferred term alphabetically within System Organ Class.

Table 112: Summary of Subjects with Adverse Events by Severity and Relationship – ASP8062

| | Number of Subjects (%) (N=x) | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Mild Moderate Severe Life-threatening All Grades | | | | | | | | | | | |
| | MedDRA | R | NR | R | NR | R | NR | R | NR | R | NR | R + NR |
| SOC | PT | | | | | | | | | | | |
| | | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |

Notes: Events are counted once per subject at the highest severity grade and closest relationship to the investigational product. R= related to investigational product (possibly, probably, definitely). NR = not related to investigational product (unrelated, unlikely).

Table 113: Summary of Subjects with Adverse Events by Severity and Relationship – Placebo

| | Number of Subjects (%) (N=x) | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Mild Moderate Severe Life-threatening All Grades | | | | | | | | | | | |
| SOC | MedDRA<br>PT | R | NR | R | NR | R | NR | R | NR | R | NR | R + NR |
| | XX | | | | | | | | | | | |

Notes: Events are counted once per subject at the highest severity grade and closest relationship to the investigational product. R= related to investigational product (possibly, probably, definitely). NR = not related to investigational product (unrelated, unlikely).

Table 114: Number and Percentage of Subjects with Adverse Events by Maximum Severity - Safety Subjects

| MedDRA SOC/ | edDRA SOC/ | | | | Placebo | | | |
|---|---|---|---|---|---|---|---|---|
| Preferred Term | | (N= | =xx) | | (N=xx) | | | |
| | | | | Life- | Li | | | |
| | Mild | Moderate | Severe | threatening | Mild | Moderate | Severe | threatening |
| - Any Adverse Events - | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| SOC | | | | | | | | |
| - Overall - | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Preferred term 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

Notes: Percentages are based on the total number of subjects, as given in the column heading.

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term.

Table 115: Number and Percentage of Subjects Adverse Events by Relatedness - Safety Subjects

| MedDRA SOC/ | ASI | P8062 | Placebo | |
|---|---|---|---|---|
| Preferred Term | (n= | =xx) | (n=x | x) |
| | Related <sup>1</sup> | Not-Related <sup>2</sup> | Related | Not-Related |
| SOC | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| - Overall - | | | | |
| Preferred term 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

<sup>&</sup>lt;sup>1</sup>Related are possibly, probably or definitely related to investigational product

<sup>&</sup>lt;sup>2</sup> Not Related to investigational product (not related or unlikely)

Table 116: Number and Percentage of Subjects with Treatment-Related Adverse Events by Maximum Severity- Safety Subjects

| MedDRA SOC/ | | ASP8062 | | | | Placebo | | |
|---|---|---|---|---|---|---|---|---|
| Preferred Term | | (N=xx) | | | | (N=xx) | | |
| | Life- | | | | | | Life- | |
| | Mild | Moderate | Severe | threatening | Mild | Moderate | Severe | threatening |
| SOC | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| - Overall - | | | | | | | | |
| Preferred term 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term.

Table 117: Number and Percentage of Subjects with Adverse Events Occurring in >= 5% of Subjects in Any One Group - Safety Subjects

| MedDRA SOC/ | ASP806 | Placebo | |
|------------------|------------|------------|----------------------|
| Preferred Term | (N=xx) | (N=xx) | p-value <sup>1</sup> |
| SOC | nn (xx.x%) | nn (xx.x%) | X.XXX |
| - Overall - | | | |
| Preferred term 1 | nn (xx.x%) | nn (xx.x%) | X.XXX |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) | x.xxx |

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term. At least % occurring in either arm to be included in the table.

Programmer's Notes: Order System Organ Class alphabetically and preferred term alphabetically within System Organ Class.

Table 118: Number and Percentage of Subjects with Adverse Events Leading to Discontinuation of Study - Safety Subjects

| MedDRA SOC/ | ASP8062 | Placebo |
|------------------|------------|------------|
| Preferred Term | (N=xx) | (N=xx) |
| SOC | | |
| - Overall - | nn (xx.x%) | nn (xx.x%) |
| Preferred term 1 | nn (xx.x%) | nn (xx.x%) |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) |

Notes: Percentages are based on the total number of subjects, as given in the column heading.

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term.

<sup>&</sup>lt;sup>1</sup>p-value from Fisher's exact test

Table 119: Number and Percentage of Subjects with Adverse Events Leading to Discontinuation of Study Drug – Safety Subjects

| MedDRA SOC/ | ASP8062 | Placebo |
|------------------|------------|------------|
| Preferred Term | (N=xx) | (N=xx) |
| SOC | | |
| - Overall - | nn (xx.x%) | nn (xx.x%) |
| Preferred term 1 | nn (xx.x%) | nn (xx.x%) |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) |

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term.

**Table 120:** CIWA-AR Score ≥ 10 at Least Once During Treatment – Safety Subjects

| | ASP8062 | Placebo | | | | 95% CI <sup>2</sup> | |
|---|---|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | p-value <sup>1</sup> | Cohen's h | Odds Ratio | OR <sup>3</sup> Lower CI | OR Upper CI |
| CIWA-AR Score >= 10 | | | | | | | |
| Never | xx (xx.x%) | xx (xx.x%) | | | | | |
| At Least Once | xx (xx.x%) | xx (xx.x%) | 0.xxx | | | | |
| ASP8062 vs Placebo | | | | 0.xx | XX.XXX | XX.XXX | XX.XXX |

1 Chi-squared test; <sup>2</sup> CI is confidence interval; <sup>3</sup> OR is odds ratio

Table 121: Summary of Vital Signs and Body Weights – Safety Subjects

| | | ASP8062 | | | | | Placebo | |
|---|---|---|---|---|---|---|---|---|
| Parameter | N | Mean (SD) | Med | Min-Max | N | Mean (SD) | Med | Min-Max |
| Vital Sign (units) | | | | | | | | |
| Screening | XX | xx.x (xx.xx) | XX.X | (xx.x - xx.x) | XX | xx.x (xx.xx) | XX.X | (xx.x - xx.x) |
| Week 1 | XX | xx.x (xx.xx) | XX.X | (xx.x - xx.x) | XX | xx.x (xx.xx) | XX.X | (xx.x - xx.x) |
| Change from Baseline | XX | xx.x (xx.xx) | XX.X | (xx.x - xx.x) | XX | xx.x (xx.xx) | XX.X | (xx.x - xx.x) |
| Weeks 2,3,4,5,6,7 | | | • | | | | | |

Programmers note: vital signs include pulse rate, systolic blood pressure, and diastolic blood pressure. Body weight (kg) will also be presented.

**Table 122:** Summary of ECG Results - Safety Subjects

| | ASP8062 | Placebo |
|--------------------------------------|------------|------------|
| Result | (N=xx) | (N=xx) |
| Screening | | |
| Normal | nn (xx.x%) | nn (xx.x%) |
| Abnormal, Not Clinically Significant | nn (xx.x%) | nn (xx.x%) |

| Abnormal, Clinically Significant | nn (xx.x%) | nn (xx.x%) |
|--------------------------------------|------------|------------|
| Week 4 | | |
| Normal | nn (xx.x%) | nn (xx.x%) |
| Abnormal, Not Clinically Significant | nn (xx.x%) | nn (xx.x%) |
| Abnormal, Clinically Significant | nn (xx.x%) | nn (xx.x%) |
| Week 7 | | |
| Normal | nn (xx.x%) | nn (xx.x%) |
| Abnormal, Not Clinically Significant | nn (xx.x%) | nn (xx.x%) |
| Abnormal, Clinically Significant | nn (xx.x%) | nn (xx.x%) |

Table 123: Summary of Blood Chemistries and Hematology – Safety Subjects

| | ASP8062 | | | | Placebo | | | |
|---|---|---|---|---|---|---|---|---|
| | N | Mean (SD) | Med | (Min-Max) | N | Mean (SD) | Med | (Min-Max) |
| Chemistry (units) | | | | | | | | |
| Baseline Value | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | XX | xx.x (xx.x) | xx.x | (xx.x-xx.x) |
| Week 4 | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) |
| Change from baseline | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) |
| Week 7 | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) |
| Change from baseline | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) |

Programmers note: table will include creatinine, ALT, AST, total bilirubin, alkaline phosphate, albumin, CrCl, GGT, RBC, WBC, hematocrit, hemoglobin, platelets.

**Table 124:** Summary of Urinalysis Continuous Data – Safety Subjects

| ASP8062 | Placebo |
|---------|---------|
|---------|---------|

| | N | Mean (SD) | Med | (Min-Max) | N | Mean (SD) | Med | (Min-Max) |
|---|---|---|---|---|---|---|---|---|
| Urinalysis (units) | | | | | | | | |
| Baseline Value | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) |
| Week 4 | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) |
| Change from baseline | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) |
| Week 7 | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) |
| Change from baseline | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) |

Programmers note: table will PH, specific gravity, and glucose result, .

**Table 125:** Summary of Urine Glucose and Nitrites – Safety Subjects

| | ASP | 8062 | Placebo | | |
|----------|-----------|-----------|-----------|-----------|--|
| | Positive | Negative | Positive | Negative | |
| | n (%) | n (%) | n (%) | n (%) | |
| Glucose | | | | | |
| Baseline | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Week 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Week 7 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Nitrites | | | | | |
| Baseline | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
|----------|-----------|-----------|-----------|-----------|
| Week 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Week 7 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Table 126: Summary of Urine Protein, Ketones, Billirubin, Leukocyte Esterace, and Blood – Safety Subjects

| | | ASP8062 | | | Placebo | |
|---|---|---|---|---|---|---|
| | Baseline | Baseline Week 4 Week 7 | | Baseline | Week 4 | Week 7 |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Blood | | | | | | |
| Negative | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Trace | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ketones | | | | | | |
| Negative | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

| Trace | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
|---|---|---|---|---|---|---|
| 1+ (small) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2+ (medium) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3+ (large) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protein | | | | | | |
| Negative | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Trace | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Programmer Note: Billirubin and Leukocyte Esterace follow the same as Protein

Table 127: Summary of Positive Urine Drug Tests, Preganancy Test or BAC > 0.02 Any Time During the Study– Safety Subjects

| Test | ASP8062 | Placebo |
|------|---------|---------|
|------|---------|---------|

| | (N=xx) | (N=xx) |
|------------------------|----------|----------|
| THC | xx (xx%) | xx (xx%) |
| Cocaine | xx (xx%) | xx (xx%) |
| Opioids | xx (xx%) | xx (xx%) |
| Methamphetamine | xx (xx%) | xx (xx%) |
| Amphetamine | xx (xx%) | xx (xx%) |
| MDMA | xx (xx%) | xx (xx%) |
| Benzodiazapines | xx (xx%) | xx (xx%) |
| Buprenorphine | xx (xx%) | xx (xx%) |
| Methadone | xx (xx%) | xx (xx%) |
| Oxycodone | xx (xx%) | xx (xx%) |
| Ethylglucuronide (EtG) | xx (xx%) | xx (xx%) |
| Pregnancy | xx (xx%) | xx (xx%) |
| BAC > 0.02 | xx (xx%) | xx (xx%) |

Table 128: Frequency of Subjects with Suicidal Ideation Any Time During the Study – Safety Subjects

| ASP8062 | Placebo | p-value |
|------------|------------|---------|
| (N=xx) | (N=xx) | |
| xx (xx.x%) | xx (xx.x%) | 0.xxx |

**Table 129:** Return to Baseline ACQ-SF-R Scores – Safety Subjects

| | ASP8062 | Placebo |
|--------------------------|----------|----------|
| Test | (N=xx) | (N=xx) |
| Screening | | |
| Increased Craving, n (%) | xx (xx%) | xx (xx%) |
| Week 3 | | |
| Increased Craving, n (%) | xx (xx%) | xx (xx%) |

# 12.2. Listings

**Listing 1: Subject Disposition - All Subjects** 

| Subject<br>ID | Date of<br>Consent | Treatment<br>Group | mITT | Eval-<br>uable | Safety | Study<br>Completion | (Day) Date of<br>Study<br>Completion or<br>Early<br>Withdrawal | Reason for Early<br>Withdrawal | Subject<br>confined | Start Date/ End<br>Date of<br>confinement |
|---|---|---|---|---|---|---|---|---|---|---|
| xxx | ddmmmyyyy | ASP8062 | Yes | Yes | Yes | Yes | (xx) ddmmmyyyy | xxxxxx | Yes | ddmmmyyyy /<br>ddmmmyyyy |
| | | Placebo | No | No | No | No | | | No | |
| | | None | | | | | | | | |

Note: Day is relative to Study Day 0.

Listing 2. Enrollment and Randomization – All Consented Subjects

| Subject ID | Treatment Group | Did the subject meet all eligibility criteria? | Randomized? | Date of Randomization | Kit Number |
|---|---|---|---|---|---|
| XXX | ASP8062 | Yes | Yes | ddmmmyyyy | XXX |
| | Placebo | No | No | | |

**Listing 3: Reason not Eligible – Screen Failures** 

| Subject ID | Criterion Type | Criterion |
|------------|--------------------|-----------|
| XXX | Inclusion Criteria | |
| | Exclusion Criteria | |

**Listing 4: Protocol Deviations – Safety Subjects** 

| Subject ID | Treatment Group | <b>Deviation Date</b> | Protocol Deviation | Details |
|---|---|---|---|---|
| | | | Subject Failed to Meet the Inclusion/Exclusion | |
| XXX | ASP8062 | ddmmmyyyy | Criteria | |
| | Placebo | | Source Documentation was Not Available | |
| | | | Pregnancy Test Not Performed | |
| | | | Required study data was not obtained or obtained | |

| late due to site error | |
|----------------------------|---------------|
| Informed Consent Deviation | |
| AE/SAE Reporting Deviation | |
| Other Deviation: | xxxxxxxxxxxxx |

Note: Only subjects with protocol deviation are listed.

Listing 5: Subjects Excluded from the Efficacy Analysis or Evaluable Set

| Subject<br>ID | Treatment Group | Reason for Exclusion from mITT | Reason for Exclusion from Evaluable Set |
|---|---|---|---|
| XXX | ASP8062 | XXXXXX | |
| | Placebo | | |

Note: Only subjects excluded from the efficacy analysis or evaluable set are listed.

**Listing 6: Demographics Data – Safety Subjects** 

| Subject<br>ID | Treatment Group Gender Age (yrs) E | | Ethnicity | Race | |
|---|---|---|---|---|---|
| xxx | ASP8062 | Male | XX | Hispanic or Latino | American Indian or Alaska<br>Native |
| | Placebo | Female | | Not Hispanic or Latino | Asian |
| | | | | Unknown | Native Hawaiian or Other<br>Pacific Islander |
| | | | | | Black or African American |
| | | | | | White |
| | | | | | Other |
| | | | | | Unknown |

**Listing 7: Baseline Drinking Characteristics – mITT Subjects** 

| Subject<br>ID | Treatment<br>Group | Drinks/Day<br>(Days -1 to -28) | Drinks/Day<br>(Days -1 to -14<br>Pre-<br>randomization) | Drinks/ Drinking<br>Day<br>(Days -1 to -28) | Drinks/Drinking<br>Day (Days -1 to -14<br>Pre-randomization) | Weekly % Heavy<br>Drinking Days<br>(Days -1 to -28) | Weekly % Heavy Drinking Days (Days -1 to -14 Pre- randomization) |
|---|---|---|---|---|---|---|---|
| XXX | ASP8062 | XXX.X | XXX.X | xxxx | XXX.X | XXX.X | XXX.X |
| | Placebo | | | | | | |

| Subject | Treatment | Weekly %Very | Weekly % Very | Weekly % Days | Weekly % Days |
|---|---|---|---|---|---|
| Bublect | 11 Catillett | VICCINITY /UVCITY | VICCINIY /U VCI y | WCCKIY /U Days | WCCKIY /U Days |

| ID | Group | Heavy Drinking<br>Days<br>(Days -1 to -28) | Heavy Drinking<br>Days<br>(Days -1 to -14 Pre-<br>randomization) | Abstinent<br>(Days -1 to -28) | Abstinent (Days -1<br>to -14 Pre-<br>randomization) |
|---|---|---|---|---|---|
| XXX | ASP8062 | XXX.X | XXX.X | XXX.X | XXX.X |
| | Placebo | | | | |

Note: Exclude the three abstinent days during pre-randomization period.

**Listing 8: Baseline Smoking Characteristics – mITT Subjects** 

| Subject ID | Treatment Group | Over the past week, how many days did you smoke cigarettes? | How many cigarettes on average per day? | Over the past week, how many days did you use nicotine products? |
|---|---|---|---|---|
| xxx | ASP8062 | None | XXX | None |
| | Placebo | 1, 2, 3, 4, 5 | | 1, 2, 3, 4, 5 |
| | | 6, 7 | | 6, 7 |
| | | Refused to answer | | Refused to answer |

**Listing 9: MINI DSM-5 Disorders – Safety Subjects** 

| Subject<br>ID | Treatment Group | Visit Date | Diagnosis | Timeframe |
|---------------|-----------------|------------|-----------|-------------------|
| XXX | ASP8062 | ddmmmyyyy | xxxxxx | Current (2 weeks) |
| | Placebo | | | Past |
| | | | | Recurrent |

Note: Only subjects with a diagnosis of a disorder will be listed.

Listing 10: MINI DSM-5 AUD – Safety Subjects

| Subject<br>ID | Treatment<br>Group | Visit Date | # of Symptoms |
|---------------|--------------------|------------|---------------|
| XXX | ASP8062 | ddmmmyyyy | XX |
| | Placebo | | |

**Listing 11: Medical History – Safety Subjects** 

| Subject<br>ID | Treatment Group | Medical History<br>Verbatim Term/<br>Preferred Term/<br>SOC | Start Date | Ongoing |
|---|---|---|---|---|
| XXX | ASP8062 | xxxxxxxxxx | ddmmmyyyy | No |
| XXX | | xxxxxxxxxx | ddmmmyyyy | |

Programming note: Only identify items that were scored "yes"

**Listing 12: Drinking Goal – mITT Subjects** 

| Subject<br>ID | Treatment<br>Group | Visit Date | Time | What goal have you chosen for yourself about drinking by the end of the study? | What might a typical week look like at the end of the study having achieved your goal? (number of drinks per day) | Motivation to reach goal | Confidence to reach goal |
|---|---|---|---|---|---|---|---|
| XXX | ASP8062 | ddmmmyyyy | hh:mm | To stop drinking | XX | XX | XX |
| | Placebo | | | Reduce drinking but not stop | | | |

**Listing 13: Physical Exam – Safety Subjects** 

| Subject<br>ID | Treatment Group | Exam Date | Finding | Any abnormal finding during the physical exam? |
|---|---|---|---|---|
| XXX | ASP8062 | ddmmmyyyy | XXXXXXXXXX | Yes |
| | Placebo | | | No |

Programming Note: Only report the items that are abnormal

Listing 14: Daily and Weekly Standard Drink Units (TLFB) During Treatment – mITT Subjects

| Subject<br>ID | Treatment<br>Group | Week | D1 | D2 | D3 | <b>D4</b> | D5 | D6 | <b>D7</b> | Mean<br>drinks/day | Mean drinks/<br>drinking day | Heavy<br>drinking days | % days<br>abstinent |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX | ASP8062 | 1 | XX | XX | XX | XX | XX | XX | XX | | | | |
| | Placebo | 2 | | | | | | | | | | | |
| | | 3, etc | | | | | | | | | | | |

## **Listing 15: Brief Drinking Questionnaire – mITT Subjects**

| Subject<br>ID | Treatment<br>Group | Date of<br>Assessment | Date that the last day of non-<br>missing drinking data was<br>collected by TLFB | This is a period of XX days since the last day of drinking data that was collected by TLFB | Did the subject drink during this period? | How many days during this period did the subject drink? |
|---|---|---|---|---|---|---|
| XXX | ASP8062 | ddmmmyyyy | ddmmmyyyy | xx | Yes | XX |
| | Placebo | | | | No | |

| | | | How many | | Maximum number of | How many days did you |
|---|---|---|---|---|---|---|
| Subject | Treatment | Date of | alcoholic drinks | How many heavy | drinks on any one | drink this maximum |
| ID | Group | Assessment | on a typical day? | drinking days? | day? | number? |
| XXX | ASP8062 | ddmmmyyyy | XX | XX | XX | XX |
| | Placebo | | | | | |

# **Listing 16: Cue Reactivity – mITT Subjects**

| Subject<br>ID | Treatment<br>Group | Visit | Date of<br>Assessment | Assessment<br>Time | Cue | How strong is your craving to drink alcohol? | Having a drink<br>would make things<br>just perfect | If I could drink<br>alcohol now, I<br>would drink it |
|---|---|---|---|---|---|---|---|---|
| xxx | ASP8062 | Screening | ddmmmyyyy | hh:mm | Water | xx | xx | xx |

| PI | Placebo | Week 2 | Alcohol |
|-------|---------|--------|---------|
| 1 1 1 | laccoo | | |

| Subject<br>ID | Treatment<br>Group | Visit | Cue | It would be hard<br>to turn down a<br>drink right now | How much did<br>you like the<br>beverage just<br>given to you? | Sum of first 4 questions |
|---|---|---|---|---|---|---|
| xxx | ASP8062 | Screening | Water | xx | xx | xx |
| | Placebo | Week 2 | Alcohol | | | |

# **Listing 17: Drinking Consequences and Craving Scores – mITT Subjects**

| | | | | | | | | Hyperkatifeia | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Treatment<br>Group | Week | CIWA-<br>AR | ACQ-SF-R<br>Pre | ACQ-SF-R<br>Post | PACS | PROMIS<br>Negative<br>Consequences | Total | Stress | Depress<br>ion | Irritable | Pain |
| XXX | ASP8062 | | XXX | XXX | XXX | XXX | XXX | XXX | | | | |
| | Placebo | | | | | | | | | | | |

# **Listing 18: Pittsburg Sleep Quality Index Scores – mITT Subjects**

| Subject ID | Treatment Group | Week | Total score |
|------------|-----------------|-----------|-------------|
| XXX | ASP8062 | Screening | XX |
| | Placebo | Week 6 | |

| Week 7 |
|--------|

**Listing 19: Smoking and Other Nicotine Use Data-mITT Subjects** 

| Subject<br>ID | Treatment Group | Week | Visit Date | Over the past<br>week, how many<br>days did you<br>smoke cigarettes? | On the days you<br>smoked, how<br>many cigarettes<br>did you smoke on<br>average? | How many days use nicotine products during the past week? |
|---|---|---|---|---|---|---|
| XXX | ASP8062 | | ddmmmyyyy | X | XX | X |
| | Placebo | | | | | |

**Listing 20: MINI AUD- Safety Subjects** 

| Subject | Treatment | | | | | | | | | | | | # of Symptoms |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | Group | | | | | | Item | | | | | | |
| | | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | |
| XXX | ASP8062 | Y | Y | Y | Y | Y | Y | Y | Y | Y | Y | Y | |
| | Placebo | N | N | N | N | N | N | N | N | N | N | N | |
| | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | |

| Item # | List of Items |
|---|---|
| 1 | a. During the times when you drank alcohol, did you end up drinking more than you planned when you started? |
| 2 | b. Did you repeatedly want to reduce or control your alcohol use? Did you try to cut down or control your alcohol use, but failed? IF YES TO EITHER, MARK YES. |
| 3 | c. On the days that you drank, did you spend substantial time obtaining alcohol, drinking, or recovering from the effects of alcohol? |
| 4 | d. Did you crave or have a strong desire or urge to use alcohol? |
| 5 | e. Did you spend less time meeting your responsibilities at work, at school, or at home, because of your repeated drinking? |
| 6 | f. If your drinking caused problems with your family or other people, did you still keep on drinking? |
| 7 | g. Were you intoxicated more than once in any situation where you or others were physically at risk, for example, driving a car, riding a motorbike, using machinery, boating, etc.? |
| 8 | h. Did you continue to use alcohol, even though it was clear that the alcohol had caused or worsened psychological or physical problems? |
| 9 | i. Did you reduce or give up important work, social or recreational activities because of your drinking? |
| 10 | j. Did you need to drink a lot more in order to get the same effect that you got when you first started drinking or did you get much less effect with continued use of the same amount? |
| 11 | K1. When you cut down on heavy or prolonged drinking did you have any of the following: [increased sweating or heart rate; hand tremor or "the shakes"; trouble sleeping; nausea or vomiting; hearing or seeing things other people could not see or hear or having sensations in your skin for no apparent reason; agitation; anxiety; seizures] (If yes to 2 or more of these, check yes for this question), OR K2. Did you drink alcohol to reduce or avoid withdrawal symptoms or to avoid being hung over? If K1 or K2 = yes, then score as yes. |

**Listing 21. Exit Interview – mITT Subjects** 

| Subject<br>ID | Treatment<br>Group | Visit Date | Did you think you were receiving the study drug or the placebo? | What is your desire to please people? | If you had the opportunity in the future to take the study drug again, would you continue to take it for more than 5 weeks? | Did you limit your drinking<br>because of flushing (a heat<br>reaction or facial redness)? |
|---|---|---|---|---|---|---|
| XXX | ASP8062 | ddmmmyyyy | Placebo | More than average | Yes | Yes |
| | Placebo | | Study Drug | Average | No | No |
| | | | Don't know | Less than average | Refuse to answer | Refuse to answer |
| | | | Refuse to answer | Refuse to answer | | |

| Subject<br>ID | Treatment<br>Group | Visit Date | Did you limit<br>your drinking<br>because of nausea<br>or other effects? | Did your<br>friends or<br>family notice<br>flushing? | If your friends or family noticed flushing, did this change your drinking? | Did you ever miss<br>a dose of<br>medication to<br>avoid these<br>effects? | Did you use any other services during the study to help you reduce drinking? |
|---|---|---|---|---|---|---|---|
| XXX | ASP8062 | ddmmmyyyy | Yes | Yes | Yes | Yes | Yes |
| | Placebo | | No | No | No | No | No |
| | | | | Refuse to | | | |
| | | | Refuse to answer | answer | Refuse to answer | Refuse to answer | Refuse to answer |

**Listing 22: Drug Exposure from AiCure- mITT Subjects** 

| Subject<br>ID | Treatment<br>Group | Study<br>Week | Day 1 | Day 2 | Day 3 | Day 4 | Day 5 | Day 6 | Day 7 | Total<br>Taken | Total<br>Expected |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX | • | 1, 2, 3, 4, | x | X | X | X | X | X | X | XX | XX |
| | ASP8062 | 5,6 | | | | | | | | | |
| | Placebo | | | | | | | | | | |

# **Listing 23: Drug Accountability – Safety Subjects**

| Subject ID | Treatment Group | Blister Pack | Date Dispensed | Date Returned | # Pills Returned |
|---|---|---|---|---|---|
| xxx | ASP8062 | 1, 2, 3, 4 | ddmmmyyyy | ddmmmyyyy | xx |
| | Placebo | | | | |

## **Listing 24: Take Control – mITT Subjects**

| Dates Modules Viewed |
|----------------------|
|----------------------|

| Subject<br>ID | Treatment Group | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
|---|---|---|---|---|---|---|---|---|
| xxx | ASP8062 | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy |
| | Placebo | | | | | | | |

**Listing 25: Adverse Events – Safety Subjects** 

| Subject<br>ID | Treatment<br>Group | Adverse Event<br>(Verbatim) S:<br>SOC<br>P: PT<br>Term | Start Date/<br>Day | Stop Date/<br>Day | Duration<br>in Days | Severity | Relation<br>-ship | Actions<br>Taken | Outcome | Serious |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | ddmmmyyyy/ | ddmmmyyyy/ | | | | | | |
| XXX | ASP8062 | Verbatim | XX | XX | | 1 | 1 | 1 | 1 | Yes |
| | Placebo | S: xxxx | XX | XX | | 2 | 2 | 2 | 2 | No |
| | | P: xxxx | | | | 3 | 3 | 3 | 3 | |
| | | | | | | 4 | 4 | 4 | 4 | |
| | | | | | | | 5 | 5 | 5 | |
| | | | | | | | | 6 | | |

Notes: Day is relative to Study Day 0.

Severity: 1=Mild; 2=Moderate; 3=Severe; 4=Potentially Life-threatening. Relationship: 1= Unrelated; 2=Unlikely; 3=Possibly; 4=Probably; 5=Definitely

Action Taken Due to AE: 1=None; 2=Treated with Drugs; 3=Non-drug treatment; 4=ER/Outpatient visit; 5=Hospitalization; 6=Referral for treatment

Outcome: 1=Resolved; 2=Recovered with sequelae; 3=Ongoing; 4=Required treatment; 5=Unknown

Programmer's Note: If "Were any AEs reported?" checkbox=No, then display "None Reported" in the Adverse Event column and SOC/PT column. If an AE started and stopped the same day, the duration is 1 day.

**Listing 26: Serious Adverse Events – Safety Subjects** 

| Subject | Treatment | SAE<br>Verbatim<br>S: SOC | Start Date/ | Stop Date/ | | SAE | Relevant<br>tests/<br>laboratory |
|---|---|---|---|---|---|---|---|
| ID | Group | P: PT | Day | Day | SAE Category | Description | data |
| XXX | ASP8062 | Verbatim | ddmmmyyyy | ddmmmyyyy | Results in Death | | XXXXXX |
| | Placebo | S: XXX | Xx | Xx | Life-threatening | | |

| | Requires or Prolongs |
|-------|----------------------------------|
| P: XX | Hospitalization |
| | Disability |
| | Congenital Anomaly/Birth |
| | Defect |
| | Required Intervention to Prevent |
| | Persistant or Significant |
| | Disability / Incapacity |
| | Other |

| Subject<br>ID | SAE | Date of death | Cause of death | Hospitalization<br>Date/Discharge<br>Date | Comments |
|---|---|---|---|---|---|
| XXX | Verbatim | ddmmmyyyy | XXXXXX | ddmmmyyyy | xxxxxxxxxxxxxxxxx |
| | | | | ddmmmyyyy | |

Notes: Day is relative to Study Day 0.

Severity: 1=Mild; 2=Moderate; 3=Severe; 4=Potentially Life-threatening. Relationship: 1= Unrelated; 2=Unlikely; 3=Possibly; 4=Probably; 5=Definitely

Outcome: 1=Recovered/Resolved; 2=Recovering/Resolving; 3=Not Recovered/Not Resolved; 4=Recovered/Resolved With Sequelae; 5=Fatal (Date of Death)

**Listing 27: POMS Scores – mITT Subjects** 

| | | | | Scores | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Treatment<br>Group | Week | Total Mood<br>Disturbance | Tension | Depression | Anger | Fatigue | Confusion | Vigor |
| XXX | ASP8062 | | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| | Placebo | | | | | | | | |

Listing 28. Columbia-Suicide Severity Scale – Safety Subjects

| | | | | Response | Response to Question: | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Treatment<br>Group | Visit Date | Study<br>Week | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 | Q7 | Q8 | Q9 | Q10 | Q11 | Q12 | Q13 |
| XXX | ASP8062 | ddmmmyyyy | | Yes | Yes | Yes | Yes | Yes | Yes | Type 1 | 1 | 1 | 0 | 0 | 0 | Yes |
| | Placebo | | | No | No | No | No | No | No | Type 2 | 2 | 2 | 1 | 1 | 1 | No |
| | | | | | | | | | | Type 3 | 3 | 3 | 2 | 2 | 2 | |
| | | | | | | | | | | Type 4 | 4 | 4 | 3 | 3 | 3 | |
| | | | | | | | | | | Type 5 | 5 | 5 | 4 | 4 | 4 | |
| | | | | | | | | | | | | | 5 | 5 | 5 | |

#### Suicide Ideation

- 1. Have you wished you were dead or wished you could go to sleep and not wake up?
- 2. Have you actually had any thoughts of killing yourself?
- 3. Have you been thinking about how you might do this?
- 4. Have you had these thoughts and had some intention of acting on them?
- 5. Have you started to work out or worked out the details of how to kill yourself?
- 6. Do you intend to carry out this plan?

#### **Intensity of Ideation**

- 7. The following features should be rated with respect to the most severe type of ideation (i.e. 1-5 with 1 being the least severe and 5 being the most severe)
- 8. How many times have you had these thoughts?1=Less than once a week; 2=Once a week; 3=2-5 times a week; 4=Daily or almost; 5=Many times each day
- 9. When you have the thoughts, how long do they last? 1=Fleeting-few seconds or minutes; 2=Less than 1 hr-some of the time; 3=1-4 hrs/a lot of time; 4=4-8 hrs/most of day; 5=More than 8 hours/persistent or continuous
- 10. Could/can you stop thining about killing yourself or wanting to die if you want to? 1=Easily; 2=Little Difficulty; 3=Some Difficulty; 4=Lot of Difficulty; 5=Unable to control; 0=Does not attempt to control
- 11. Are there things that stop you from wanting to die or acting on thoughts of committing suicide? 1=Definite deterrents; 2=Probably Deterrents; 3=Uncertain Deterrents; 4=Unlikely Deterrents; 5=No Deterrents; 0=Does not apply
- 12. What sort of reasons did you have for thinking about wanting to die or killing yourself? Was it to end pain or stop the way you were feeling or to get attention, revenge or reaction from others 1=Completely to get attention or revenge or reaction; 2=Mostly to get attention or revenge or reaction; 3=Equally to get attention or revenge or reaction and stop pain; 4=Mostly to stop pain; 5=Completely to stop pain; 0=Does not apply

#### **Suicidal Behavior**

13. Have you made a suicide attempt?

| | | | Respons | e to Quest | ion: | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Treatment<br>Group | Study<br>Week | Q14 | Q15 | Q16 | Q17 | Q18 | Q19 | Q20 | Q21 | Q22 | Q23 | Q24 |
| XXX | ASP8062 | | XX | Yes | Yes | XX | Yes | XX | Yes | Yes | Yes | 0 | 0 |
| | Placebo | | | No | No | | No | | No | No | No | 1 | 1 |
| | | | | | | | | | | | | 2 | 2 |
| | | | | | | | | | | | | 3 | |
| | | | | | | | | | | | | 4 | |
| | | | | | | | | | | | | 5 (date ddmmmyyyy) | |

- 14. Number of attempts
- 15. Has the subject engaged in non-suicidal self-injurious behavior?
- 16. Has there been a time when you started to do something to end your life but someone or something stopped you before actually did anything?
- 17. Number interrupted
- 18. Has there been a time when you stared to do something to try to end your life but you stopped yourself before you actually did anything?
- 19. Number aborted
- 20. Have you taken any step towards making a suicide attempt or preparing to kill yourself?
- 21. Suicidal behavior was present during the assessment period
- 22. Completed suicide?
- 23. Actual Lethality/Medical Damage; 0=No physical damage; 1=Minor physical damage; 2=Moderate physical Damage; 3=Moderately severe physical damage; 4=Severe physical damage; 5=Death
- 24. Potential Lethality; 0=Behavior not likely to result in injury; 1=Behavior likely to result in injury, but not death; 2=Behavior likely to result in death

## **Listing 29: Blood Chemistries – Safety Subjects**

| Subject<br>ID | Treatment Group | Visit Date | Test Name | Result | Units | Flag | Evaluation |
|---|---|---|---|---|---|---|---|
| XXXX | ASP8062 | ddmmmyyyy | Creatinine | x.xx | mg/dL | H (high) | WNL |
| | Placebo | | Total Bilirubin | XXX | mg/dL | L (low) | Abnormal, NCS |
| | | | ALT | XX.X | U/L | | Abnormal, CS |
| | | | AST | x.xx | U/L | | |
| | | | BUN | Xx | mg/dL | | |
| | | | Creatinine Clearance | XXX.XX | mL/min | | |
| | | | Akaline Phosphate | XXX.X | U/L | | |

| Subject<br>ID | Treatment Group | Visit Date | Test Name | Result | Units | Flag | Evaluation |
|---|---|---|---|---|---|---|---|
| | | | Albumin | XX.X | g/dL | | |
| | | | GGT | XX.X | U/L | | |
| | | | Total Cholesterol | XXX | mg/dL | | |
| | | | Triglycerides | XX | mg/dL | | |
| | | | Chloride | XXX | mmol/L | | |
| | | | Sodium | XXX | mmol/L | _ | |
| | | | Potasium | XX.X | mmol/L | _ | |

**Listing 30: Hematology – Safety Subjects** 

| Subject<br>ID | Treatment<br>Group | Visit Date | Test Name | Result | Units |
|---|---|---|---|---|---|
| xxxx | ASP8062 | ddmmmyyyy | Hematocrit | xxx.xx | % |
| | Placebo | | Hemoglobin | xxx | g/dL |
| | | | RBC | xx.x | mil/uL |
| | | | WBC | x.xx | thous/uL |
| | | | Platelets | xxx.xx | thous/uL |
| | | | Neutrophils | xxx.x | % |
| | | | Monocytes | xx.x | % |
| | | | Eosinophils | xx.x | % |

| Subject<br>ID | Treatment<br>Group | Visit Date | Test Name | Result | Units |
|---------------|--------------------|------------|-----------|--------|-------|
| | | | Basophils | xx.x | % |

**Listing 31: Urinalysis – Safety Subjects** 

| Subject<br>ID | Treatment<br>Group | Visit Date | Study<br>Week | рН | Specific<br>Gravity | Glucose | Glucose<br>Result<br>(mg/dL) | Protein | Ketones | Blood | Nitrites | Bilirubin | Leukocyte<br>Esterase |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxx | ASP8062 | ddmmmyyyy | Screen | xx.x | x.xxx | Negative | xxxx | Negative | Negative | Negative | Negative | Negative | Negative |
| | Placebo | | x | | | Positive | | Trace | Trace | Trace | Positive | Trace | Trace |
| | | | | | | | | 1+ | 1+ | 1+ | | 1+ | 1+ |
| | | | | | | | | 2+ | 2+ | 2+ | | 2+ | 2+ |
| | | | | | | | | 3+ | 3+ | 3+ | | 3+ | 3+ |
| | | | | | | | | 4+ | 4+ | 4+ | | 4+ | 4+ |

Listing 32: Urinalysis Microscopy<sup>1</sup> – Safety Subjects

| Subject<br>ID | Treatment<br>Group | Visit Date | Test Name | Result (cells/HPF) |
|---|---|---|---|---|
| xxxx | ASP8062 | ddmmmyyyy | Microscopic RBC | xx |
| | Placebo | | Microscopic WBC | xx |
| | | | Epithelial Cells | xx |
| | | | Hyaline Casts | xx |

<sup>&</sup>lt;sup>1</sup>Only subjects that had microscopy

Listing 33: Pregnancy Test/Birth Control Data – Safety Subjects

| Subject<br>ID | Treatment Group | Gender | Pregnancy Test<br>Performed? | Pregnancy Test /<br>Visit Date | Pregnancy Result | Methods of birth control |
|---|---|---|---|---|---|---|
| XXX | ASP8062 | Male | Not Done | ddmmmyyyy | Negative | Oral Contraceptive |
| | Placebo | Female | Yes | | Positive | Vasectomy |
| | | | | | | Contraceptive Skin Patch |
| | | | | | | Intrauterine |
| | | | | | | Medroxyprogesterone |
| | | | | | | Complete Abstinence |
| | | | | | | Tubal Ligation or Postemopausal |
| | | | | | | Other: xxxxxxxxxxxxxxx |

Programming note: Only indicate birth control methods that were indicated as Yes

**Listing 34: Blood Alcohol Concentration – Safety Subjects** 

| Subject<br>ID | Treatment<br>Group | Visit Date | Study<br>Week | BAC<br>Performed | Time of BAC | BAC % |
|---|---|---|---|---|---|---|
| XXX | ASP8062 | ddmmmyyyy | X | Done | hh:mm | X.XXX |
| | Placebo | | | Not Done | | |

**Listing 35. Urine Drug Screen – Safety Subjects** 

| Subject ID | Treatment<br>Group | Visit Date | Study<br>Week | AMP <sup>1</sup> | Benzos <sup>2</sup> | Coc <sup>3</sup> | Bup <sup>4</sup> | Meth <sup>5</sup> | Methadone | Opioids | тнс | Barb <sup>6</sup> | MDMA | EtG <sup>7</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxx | ASP8062 | ddmmmyyyy | Screen | Neg | Neg | Neg | Neg | Neg | Neg | Neg | Neg | Neg | Neg | Neg |
| | Placebo | | X | Pos | Pos | Pos | Pos | Pos | Pos | Pos | Pos | Pos | Pos | Pos |

<sup>&</sup>lt;sup>1</sup>AMP = Amphetamine; <sup>2</sup>Benzos = Benzodiazapines; <sup>3</sup> Coc = Cocaine; <sup>4</sup> Bup = Buprenorphine; <sup>5</sup> Methamphetamine; <sup>6</sup>Barb = Barbituates; <sup>7</sup> EtG = Ethyl Glucuronide; Note: Neg=negative; Pos=positive

Listing 36: Vital Signs and Body Weights-Safety Subjects

| Subject ID | Treatment<br>Group | Visit Date | Study<br>Week | Weight (Kg) | Heart Rate (beats/min) | Systolic Pressure (mmHg) | Diastolic Pressure<br>(mmHg) |
|---|---|---|---|---|---|---|---|
| xxx | ASP8062 | ddmmmyyyy | Screening | XXX | XXX | XXX | XXX |
| | Placebo | | x | | | | |

## **Listing 37. ECG – Safety Subjects**

| Subject ID | Treatment Group | Visit Date | Study<br>Week | Result | If abnormal, specify finding |
|---|---|---|---|---|---|
| XXX | ASP8062 | ddmmmyyyy | Screen 1 | Normal | xxxxxxxxxx |
| | Placebo | | x | Abnormal, NCS | |
| | | | | Abnormal, CS | |

## Listing 38. Prior and Concomitant Medications – Safety Subjects

| Subject<br>ID | Treatment<br>Group | Prohibited<br>Med | Verbatin Med | Indication | Route | Frequency | Dose | Start Date/<br>Stop Date | Study Day | Continuing? |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX | ASP8062 | Yes | XXX | xxxxxx | XXXXXX | XXXXXX | XXXXXX | ddmmmyyyy | XXX | Yes |
| | Placebo | | | | | | | | | |
| | | No | XXX | | | | | | | No |

Prohibited meds include CYP3A4 inhibitors, CYP3A4 inducers, Benzodiazepines sedatives/hypnotics/anxiolytics, Monoamine oxidase inhibitors, Opioids, Opioid partial agonist-antagonists/opioid antagonists, and Drugs approved or have clinical data supporting their use for the treatment of AUD.

**Listing 39: Blood for Drug Concentrations – Safety Subjects** 

| Subject<br>ID | Treatment<br>Group | Sample<br>Collected? | Date | Time | ASP8062 Plasma<br>Level (ng/mL) | AS3486189 Plasma<br>Level (ng/mL) | AS3486191<br>Plasma Level<br>(ng/mL) | AS3486192<br>Plasma Level<br>(ng/mL) |
|---|---|---|---|---|---|---|---|---|
| xxx | ASP8062 | Yes | ddmmmyyyy | hh:mm | XXX | XXX | XXX | XXX |
| | Placebo | No | | | | | | |

**Listing 40: Comments – Safety Subjects** 

| Subject ID | Treatment Group | Comments |
|------------|-----------------|--------------|
| XXX | ASP8062 | XXXXXXXXXXXX |
| | Placebo | |

# 12.3. Figures

## Figure 1: Percentage of Subjects No Heavy Drinking Days Weeks 3-6

Programmer note: Use percent on y-axis, bar graph of PSNHDD add Cohen's h, \* a significant p-value, put values on graph

### Figure 2: Percentage of Subjects Abstinent Weeks 3-6

Programmer note: bar graph of PSA add Cohen's h, \* a significant p-value, put values on graph

## Figure 3: Weekly Percentage of Subjects No Heavy Drinking Days (mITT)

Programmer note: graph of estimates out to 5 weeks. Include 95% confidence intervals for each estimate and \* on statistically significant differences between treatment groups.

- Figure 4: Weekly Percentage of Subjects Abstinent (mITT)
- Figure 5: Weekly Percentage WHO 1-Level Decrease in Alcohol Consumption (mITT)
- Figure 6: Weekly Percentage WHO 2-Level Decrease in Alcohol Consumption No Imputation (mITT)
- Figure 7: Percentage Days Abstinent per Week Least Squares Means (mITT)
- Figure 8: Percent Heavy Drinking Days per Week Lease Squares Means –(mITT)
- Figure 9: Mean Drinks per Week Lease Squares Means (mITT)
- Figure 10: Mean Drinks per Drinking Day by Week Least Squares Means (mITT)
- Figure 11: Weekly Number of Cigarettes Smoked in Smokers Over Entire Treatment Period Least Squares Means (mITT)
- Figure 12: Clinical Chemistry, Urinalysis, and Hematology Values Over Time